CLINICAL TRIAL: NCT00772005
Title: A 24-Week, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dosage Study to Evaluate the Efficacy and Safety of Armodafinil (150, 200, and 250 mg/ Day) as Adjunctive Therapy in Adults With Schizophrenia
Brief Title: Study to Evaluate the Efficacy and Safety of Armodafinil as Adjunctive Therapy in Adults With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C10953/2034/SZ/MN
Record Dates: First submitted 2008-10-10; First posted 2008-10-15 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 150 mg/day armodafinil (Active Comparator): At the baseline visit, patients were randomly assigned to 1 of 3 armodafinil treatment groups or to the placebo treatment group. Patients took 5 tablets orally each day, once daily in the morning. Study drug was titrated (using blister cards) during the double-blind treatment period starting with 50 mg/day of armodafinil or matching placebo. The dosage of armodafinil or matching placebo tablet was increased, as applicable, by 50 mg/day on days 2, 4, 6, and 8, up to the randomized dosage of 150, 200, or 250 mg/day. Patients remained at their randomized dosage for the duration of the study.
  Interventions: Drug: armodafinil
- 200 mg/day armodafinil (Active Comparator): At the baseline visit, patients were randomly assigned to 1 of 3 armodafinil treatment groups or to the placebo treatment group. Patients took 5 tablets orally each day, once daily in the morning. Study drug was titrated (using blister cards) during the double-blind treatment period starting with 50 mg/day of armodafinil or matching placebo. The dosage of armodafinil or matching placebo tablet was increased, as applicable, by 50 mg/day on days 2, 4, 6, and 8, up to the randomized dosage of 150, 200, or 250 mg/day. Patients remained at their randomized dosage for the duration of the study.
  Interventions: Drug: armodafinil
- 250 mg/day armodafinil (Active Comparator): At the baseline visit, patients were randomly assigned to 1 of 3 armodafinil treatment groups or to the placebo treatment group. Patients took 5 tablets orally each day, once daily in the morning. Study drug was titrated (using blister cards) during the double-blind treatment period starting with 50 mg/day of armodafinil or matching placebo. The dosage of armodafinil or matching placebo tablet was increased, as applicable, by 50 mg/day on days 2, 4, 6, and 8, up to the randomized dosage of 150, 200, or 250 mg/day. Patients remained at their randomized dosage for the duration of the study.
  Interventions: Drug: armodafinil
- Matching Placebo (Placebo Comparator): At the baseline visit, patients were randomly assigned to 1 of 3 armodafinil treatment groups or to the placebo treatment group. Patients took 5 tablets orally each day, once daily in the morning. Study drug was titrated (using blister cards) during the double-blind treatment period starting with 50 mg/day of armodafinil or matching placebo. The dosage of armodafinil or matching placebo tablet was increased, as applicable, by 50 mg/day on days 2, 4, 6, and 8, up to the randomized dosage of 150, 200, or 250 mg/day. Patients remained at their randomized dosage for the duration of the study.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: armodafinil — 150 mg/day armodafinil
  Other Names: R-modafinil; CEP-10953
  Arms: 150 mg/day armodafinil
Drug: placebo — placebo
  Arms: Matching Placebo
Drug: armodafinil — 200 mg/day armodafinil
  Other Names: R-modafinil; CEP-10953
  Arms: 200 mg/day armodafinil
Drug: armodafinil — 250 mg/day armodafinil
  Other Names: R-modafinil; CEP-10953
  Arms: 250 mg/day armodafinil

SUMMARY:
The primary objective of the study is to evaluate whether armodafinil treatment is more effective than placebo as adjunctive therapy to antipsychotic medication in alleviating the negative symptoms of schizophrenia

DETAILED DESCRIPTION:
This study was designed and was powered to evaluate the efficacy and safety of armodafinil treatment at dosages of 150, 200, and 250 mg/day compared with placebo over 24 weeks as an adjunctive therapy to antipsychotic medication (olanzapine, oral risperidone, or paliperidone) in adults with schizophrenia who were clinically stable at study entry. Specifically, the effects of armodafinil treatment on the negative symptoms of schizophrenia were the primary assessment in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* The patient has a diagnosis of schizophrenia according to the DSM-IV-TR criteria and the patient has been clinically stable in a nonacute phase of their illness.
* Documentation that the patient has received treatment with olanzapine, oral risperidone, or paliperidone for schizophrenia for at least 6 weeks prior to the screening visit and has been on a stable dose of that antipsychotic medication for at least 4 weeks prior to the screening visit.
* The patient is in good health (except for the diagnosis of schizophrenia) as judged by the investigator.
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study. Acceptable methods of contraception include barrier method with spermicide, intrauterine device (IUD), steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method, or documented abstinence.
* The patient has a PANSS negative symptom score of 15 or more at the screening and baseline visits.

Key Exclusion Criteria:

* The patient has a severity rating of moderate or worse on any item of the PANSS positive symptom subscale.
* The patient has any Axis I disorder according to DSM-IV-TR criteria, including schizoaffective disorder, apart from schizophrenia and nicotine dependence, or any Axis II disorder that would interfere with the conduct of the study.
* The patient has moderate to severe depressive symptoms, as indicated by the CDSS.
* The patient has current active suicidal ideation, is at imminent risk of self-harm, or has a history of significant suicidal ideation or suicide attempt at any time in the past that causes concern at present.
* The patient has tardive dyskinesia, akathisia, moderate or worse level of extrapyramidal symptoms, or any other clinically significant movement disorder.
* The patient has a history of any cutaneous drug reaction or drug hypersensitivity reaction, a history of any clinically significant hypersensitivity reaction, or has a history of multiple clinically relevant allergies.
* The patient is a pregnant or lactating woman.
* The patient has previously received modafinil or armodafinil, or the patient has a known sensitivity to any ingredients in the study drug tablets.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (39):
- United States (39):
  - K and S Professional Research Services, LLC, Little Rock, Arkansas
  - Omega Clinical Trials, Anaheim, California
  - Synergy Clinical Research Center, Escondido, California
  - Collaborative NeuroScience, Garden Grove, California
  - Excell Research, Oceanside, California
  - CNRI Los Angeles LLC, Pico Rivera, California
  - CNRI-San Diego LLC, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Collaborative NeuroScience Network, Torrance, California
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Scientific Clinical Research, Inc., Aventura, Florida
  - Mental Health Advocates. Inc, Boca Raton, Florida
  - Fidelity Clinical Research, Lauderhill, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Comprehensive Neuroscience Inc, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Uptown Research Institute. LLC, Chicago, Illinois
  - Via Christi Research, Wichita, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Clinical Insights, Glen Burnie, Maryland
  - Sheppard Pratt Health System, Towson, Maryland
  - St Louis Clinical Trials LC, St Louis, Missouri
  - CRI Worldwide LLC, Clementon, New Jersey
  - Behavioral Medical Research of Brooklyn, Brooklyn, New York
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - Keystone Clinical Studies LLC, Norristown, Pennsylvania
  - Belmont Center for Comprehensive Treatment, Philadelphia, Pennsylvania
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Carolina Clinical Trials. Inc, Charleston, South Carolina
  - Community Clinical Research, Austin, Texas
  - FutureSearch Trials, Austin, Texas
  - University Hills Clinical Research, Irving, Texas
  - Alliance Research Group, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

REFERENCES:
- [Derived] Kane JM, Yang R, Youakim JM. Adjunctive armodafinil for negative symptoms in adults with schizophrenia: a double-blind, placebo-controlled study. Schizophr Res. 2012 Mar;135(1-3):116-22. doi: 10.1016/j.schres.2011.11.006. Epub 2011 Dec 16. PMID 22178084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 centers in the US. First participant enrolled: September 2008. Last patient completed: March 2010.
Pre-assignment Details: The study consisted of a 1- to 2-week screening period, a 24-week double-blind treatment period, and a 7-day follow-up period.
Period: Overall Study
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Started | 71 | 70 (One patient withdrew before taking any study drug.) | 72 (One patient withdrew before taking any study drug.) | 72 (Two patients withdrew before taking any study drug.)
Completed | 46 | 40 | 44 | 46
Not Completed | 25 | 30 | 28 | 26
Not completed — Adverse Event | 9 | 14 | 10 | 13
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 7 | 10 | 2
Not completed — Protocol Violation | 2 | 4 | 1 | 6
Not completed — Lost to Follow-up | 7 | 3 | 6 | 3
Not completed — Non-compliance with study procedures | 1 | 1 | 0 | 1
Not completed — Non-compliance with drug administration | 3 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo | Total
Number analyzed (Participants) | 71 | 70 | 72 | 72 | 285
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 71 | 70 | 72 | 72 | 285
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.7 (11.19) | 43.1 (11.07) | 44.4 (9.43) | 42.4 (10.07) | 43.4 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 22 | 26 | 79
  Male | 53 | 57 | 50 | 46 | 206
Region of Enrollment [Number; unit: participants]
  United States | 71 | 70 | 72 | 72 | 285

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Negative Scale Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Endpoint
Description: PANSS rates severity of psychopathology in schizophrenics. 7 items measure NEGATIVE symptoms: blunted affect, social withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Negative Scale score ranges from 7-49 (higher more severe). Data represents change in Negative Rating Scale from baseline to endpoint with positive scores indicating more severe pathology.
Time Frame: Baseline and Endpoint (Week 24 or last observation after baseline)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
Units on a scale | -2.0 (0.42) | -2.3 (0.42) | -2.1 (0.41) | -2.1 (0.42)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; Least square (LS) mean and standard error of the LS mean for each treatment group, and the p-value and 95% CI for the treatment comparisons are from an analysis of covariance (ANCOVA) with treatment as a factor and the baseline value as a covariate; Test type: Superiority or Other; p = 0.8514, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6995, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9766, ANCOVA

2. Secondary Outcome: Mean Change in Total Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Endpoint
Description: PANSS is a clinician rating severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Total scores range from 30 to 210. Data represents change in total score from baseline to endpoint, higher (positive) scores indicate more severe pathology.
Time Frame: Baseline and Endpoint (Week 24 or last observation after baseline)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
units on a scale | -3.2 (1.24) | -3.7 (1.25) | -3.4 (1.23) | -2.6 (1.25)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7596, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5620, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6688, ANCOVA

3. Secondary Outcome: Mean Change in Total Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 1
Description: PANSS rates severity of psychopathology in schizophrenics. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg.anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Total scores range from 30 to 210. The data here represents the change in total score from baseline to week 1 and higher (positive) scores indicate more severe pathology.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
Units on a scale | -1.8 (0.67) | -2.3 (0.69) | -1.0 (0.67) | -3.0 (0.67)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1894, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4582, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0327, ANCOVA

4. Secondary Outcome: Mean Change in Total Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 2
Description: PANSS is a clinician rating severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Total scores range from 30 to 210. Data represents the change in total score from baseline to week 2, higher (positive) scores indicate more severe pathology.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
Units on a scale | -4.0 (0.75) | -3.8 (0.77) | -2.0 (0.74) | -5.0 (0.75)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3275, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2597, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0039, ANCOVA

5. Secondary Outcome: Mean Change in Total Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 4
Description: PANSS is a clinician rating severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Total scores range from 30 to 210. Data represents the change in total score from baseline to week 4, higher (positive) scores indicate more severe pathology.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
Units on a scale | -4.7 (0.86) | -4.4 (0.88) | -3.6 (0.84) | -6.9 (0.86)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0713, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0431, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0063, ANCOVA

6. Secondary Outcome: Mean Change in Total Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 8
Description: PANSS is a clinician rating severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Total scores range from 30 to 210. Data represents the change in total score from baseline to week 8, higher (positive) scores indicate more severe pathology.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
Units on a scale | -4.7 (0.92) | -5.1 (0.93) | -4.7 (0.89) | -7.1 (0.91)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0619, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1137, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0598, ANCOVA

7. Secondary Outcome: Mean Change in Total Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 12
Description: PANSS is a clinician rating severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Total scores range from 30 to 210. Data represents the change in total score from baseline to week 12, higher (positive) scores indicate more severe pathology.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Units on a scale | -5.6 (1.03) | -5.2 (1.06) | -3.8 (1.02) | -6.2 (1.04)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7093, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5129, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1097, ANCOVA

8. Secondary Outcome: Mean Change in Total Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 16
Description: PANSS is a clinician rating severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Total scores range from 30 to 210. Data represent the change in total score from baseline to week 16, higher (positive) scores indicate more severe pathology.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
Units on a scale | -5.9 (1.10) | -5.5 (1.18) | -4.9 (1.11) | -7.1 (1.11)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4291, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3195, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1591, ANCOVA

9. Secondary Outcome: Mean Change in Total Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 20
Description: PANSS is a clinician rating severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Total scores range from 30 to 210. Data represents the change in total score from baseline to week 20, higher (positive) scores indicate more severe pathology.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
Units on a scale | -6.9 (1.11) | -6.0 (1.20) | -6.0 (1.16) | -7.4 (1.14)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7768, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4014, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4016, ANCOVA

10. Secondary Outcome: Mean Change in Total Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 24
Description: PANSS is a clinician rating severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Total scores range from 30 to 210. Data represent the change in total score from baseline to week 24, higher (positive) scores indicate more severe pathology.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
Units on a scale | -5.9 (1.23) | -6.8 (1.32) | -4.9 (1.25) | -6.9 (1.23)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5612, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9704, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2424, ANCOVA

11. Secondary Outcome: Mean Change in Negative Scale Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 1
Description: PANSS rates the severity of psychopathology in schizophrenics. 7 items measure negative symptoms: blunted affect, social withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Data represents change in Negative Rating Scale from baseline to week 1. Negative Scale score ranges from 7 to 49, higher (positive) score indicates more severe pathology.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
Units on a scale | -1.3 (0.27) | -0.9 (0.27) | -0.9 (0.27) | -1.3 (0.26)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8847, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2958, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2660, ANCOVA

12. Secondary Outcome: Mean Change in Negative Scale Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 2
Description: PANSS rates the severity of psychopathology in schizophrenics. 7 items measure negative symptoms: blunted affect, social withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Data represents change in Negative Rating Scale from baseline to week 2. Negative Scale score ranges from 7 to 49, higher (positive) score indicates more severe pathology.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
Units on a scale | -1.4 (0.33) | -1.3 (0.34) | -1.1 (0.33) | -2.3 (0.33)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0524, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0328, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0084, ANCOVA

13. Secondary Outcome: Mean Change in Negative Scale Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 4
Description: PANSS rates the severity of psychopathology in schizophrenics. 7 items measure negative symptoms: blunted affect, social withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Data represents change in Negative Rating Scale from baseline to week 4. Negative Scale score ranges from 7 to 49, higher (positive) score indicates more severe pathology.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
Units on a scale | -2.3 (0.37) | -1.4 (0.38) | -1.7 (0.36) | -2.8 (0.37)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3651, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0096, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0327, ANCOVA

14. Secondary Outcome: Mean Change in Negative Scale Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 8
Description: PANSS rates the severity of psychopathology in schizophrenics. 7 items measure negative symptoms: blunted affect, social withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Data represents change in Negative Rating Scale from baseline to week 8. Negative Scale score ranges from 7 to 49, higher (positive) score indicates more severe pathology.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
Units on a scale | -2.3 (0.42) | -1.9 (0.42) | -2.4 (0.40) | -3.0 (0.41)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2091, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0706, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3052, ANCOVA

15. Secondary Outcome: Mean Change in Negative Scale Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 12
Description: PANSS rates the severity of psychopathology in schizophrenics. 7 items measure negative symptoms: blunted affect, social withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Data represents change in Negative Rating Scale from baseline to week 12. Negative Scale score ranges from 7 to 49, higher (positive) score indicates more severe pathology.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Units on a scale | -2.6 (0.43) | -2.0 (0.44) | -2.5 (0.43) | -2.6 (0.43)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9960, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3604, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9528, ANCOVA

16. Secondary Outcome: Mean Change in Negative Scale Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 16
Description: PANSS rates the severity of psychopathology in schizophrenics. 7 items measure negative symptoms: blunted affect, social withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Data represents change in Negative Rating Scale from baseline to week 16. Negative Scale score ranges from 7 to 49, higher (positive) score indicates more severe pathology.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
Units on a scale | -2.9 (0.47) | -2.6 (0.50) | -2.5 (0.47) | -2.9 (0.47)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9797, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6173, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5415, ANCOVA

17. Secondary Outcome: Mean Change in Negative Scale Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 20
Description: PANSS rates the severity of psychopathology in schizophrenics. 7 items measure negative symptoms: blunted affect, social withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Data represents change in Negative Rating Scale from baseline to week 20. Negative Scale score ranges from 7 to 49, higher (positive) score indicates more severe pathology.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
Units on a scale | -3.2 (0.47) | -2.9 (0.50) | -2.8 (0.49) | -2.6 (0.48)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3547, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6642, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7395, ANCOVA

18. Secondary Outcome: Mean Change in Negative Scale Scores From the Positive and Negative Syndrome Scale (PANSS) From Baseline to Week 24
Description: PANSS rates the severity of psychopathology in schizophrenics. 7 items measure negative symptoms: blunted affect, social withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Data represents change in Negative Rating Scale from baseline to week 24. Negative Scale score ranges from 7 to 49, higher (positive) score indicates more severe pathology.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
Units on a scale | -2.5 (0.52) | -2.7 (0.56) | -2.1 (0.53) | -2.6 (0.52)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8124, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8961, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4999, ANCOVA

19. Secondary Outcome: Mean Change From Baseline to Endpoint in the Positive and Negative Syndrome Scale(PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The data here represents the change in the Positive scale score from baseline to endpoint. The scale may range from 7 to 49, higher (positive) score indicating more severe pathology.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
Units on a scale | 0.2 (3.20) | 0.2 (3.37) | -0.2 (2.78) | 0.2 (4.41)

20. Secondary Outcome: Mean Change From Baseline to Week 1 in the Positive and Negative Syndrome Scale (PANSS)Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The data here represents the change in the Positive scale score from baseline to Week 1. The scale may range from 7 to 49, higher (positive) score indicating more severe pathology.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
Units on a scale | 0.0 (1.98) | -0.4 (1.55) | -0.2 (1.59) | -0.4 (2.25)

21. Secondary Outcome: Mean Change From Baseline to Week 2 in the Positive and Negative Syndrome Scale (PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The data here represents the change in the Positive scale score from baseline to Week 2. The scale may range from 7 to 49, higher (positive) score indicating more severe pathology.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
Units on a scale | -0.6 (2.04) | -0.6 (2.04) | -0.2 (2.07) | -0.5 (1.99)

22. Secondary Outcome: Mean Change From Baseline to Week 4 in the Positive and Negative Syndrome Scale (PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The data here represents the change in the Positive scale score from baseline to Week 4. The scale may range from 7 to 49, higher (positive) score indicating more severe pathology.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
Units on a scale | -0.3 (2.30) | -0.8 (2.16) | -0.6 (2.22) | -1.2 (2.25)

23. Secondary Outcome: Mean Change From Baseline to Week 8 in the Positive and Negative Syndrome Scale (PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The data here represents the change in the Positive scale score from baseline to Week 8. The scale may range from 7 to 49, higher (positive) score indicating more severe pathology.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
Units on a scale | -0.1 (1.74) | -0.9 (2.12) | -0.7 (2.20) | -1.1 (2.31)

24. Secondary Outcome: Mean Change From Baseline to Week 12 in the Positive and Negative Syndrome Scale (PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The data here represents the change in the Positive scale score from baseline to Week 12. The scale may range from 7 to 49, higher (positive) score indicating more severe pathology.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Units on a scale | -0.5 (2.24) | -0.6 (2.75) | -0.4 (2.34) | -1.0 (2.64)

25. Secondary Outcome: Mean Change From Baseline to Week 16 in the Positive and Negative Syndrome Scale (PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The data here represents the change in the Positive scale score from baseline to Week 16. The scale may range from 7 to 49, higher (positive) score indicating more severe pathology.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
Units on a scale | -0.3 (2.62) | -0.9 (2.68) | -0.7 (2.55) | -1.2 (2.83)

26. Secondary Outcome: Mean Change From Baseline to Week 20 in the Positive and Negative Syndrome Scale (PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The data here represents the change in the Positive scale score from baseline to Week 20. The scale may range from 7 to 49, higher (positive) score indicating more severe pathology.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
Units on a scale | -0.7 (2.08) | -0.9 (2.88) | -1.0 (2.24) | -1.3 (2.42)

27. Secondary Outcome: Mean Change From Baseline to Week 24 in the Positive and Negative Syndrome Scale (PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility. Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The data here represents the change in the Positive scale score from baseline to Week 24. The scale may range from 7 to 49, higher (positive) score indicating more severe pathology.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
Units on a scale | -0.3 (2.07) | -1.0 (2.71) | -0.6 (2.36) | -1.1 (3.36)

28. Secondary Outcome: Mean Change From Baseline to Endpoint on the Positive and Negative Syndrome Scale (PANSS) General Psychopathology Scale Score
Description: PANSS rates psychopathology severity in schizophrenics. 16 items form a General Psychopathology scale:somatic concern, anxiety, guilt feeling, tension, mannerisms/posturing, depression, motor retardation, uncooperative, unusual thoughts, disorientation, poor attention, poor judgment/insight, disturbance of volition, poor impulse control, preoccupation, social avoidance. Scored on severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 16 to 112, higher (positive) score more severe pathology. Data shows change from baseline to endpoint.
Time Frame: Baseline and Endpoint (Week 24 or last observation after baseline)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
Units on a scale | -1.4 (0.68) | -1.6 (0.68) | -1.1 (0.67) | -0.7 (0.68)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4540, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3580, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6271, ANCOVA

29. Secondary Outcome: Mean Change From Baseline to Week 1 on the Positive and Negative Syndrome Scale (PANSS) General Psychopathology Scale Score
Description: PANSS rates psychopathology severity in schizophrenics. 16 items form a General Psychopathology scale:somatic concern, anxiety, guilt feeling, tension, mannerisms/posturing, depression, motor retardation, uncooperative, unusual thoughts, disorientation, poor attention, poor judgment/insight, disturbance of volition, poor impulse control, preoccupation, social avoidance. Scored on severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 16 to 112, higher (positive) score more severe pathology. Data show change from baseline to week 1.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
Units on a scale | -0.5 (0.41) | -1.0 (0.42) | 0.0 (0.41) | -1.3 (0.41)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1459, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6004, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0192, ANCOVA

30. Secondary Outcome: Mean Change From Baseline to Week 2 on the Positive and Negative Syndrome Scale (PANSS) General Psychopathology Scale Score
Description: PANSS rates psychopathology severity in schizophrenics. 16 items form a General Psychopathology scale:somatic concern, anxiety, guilt feeling, tension, mannerisms/posturing, depression, motor retardation, uncooperative, unusual thoughts, disorientation, poor attention, poor judgment/insight, disturbance of volition, poor impulse control, preoccupation, social avoidance. Scored on severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 16 to 112, higher (positive) score more severe pathology. Data show change from baseline to week 2.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
Units on a scale | -2.0 (0.43) | -2.0 (0.44) | -0.8 (0.42) | -2.1 (0.43)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8455, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8715, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0309, ANCOVA

31. Secondary Outcome: Mean Change From Baseline to Week 4 on the Positive and Negative Syndrome Scale (PANSS) General Psychopathology Scale Score
Description: PANSS rates psychopathology severity in schizophrenics. 16 items form a General Psychopathology scale:somatic concern, anxiety, guilt feeling, tension, mannerisms/posturing, depression, motor retardation, uncooperative, unusual thoughts, disorientation, poor attention, poor judgment/insight, disturbance of volition, poor impulse control, preoccupation, social avoidance. Scored on severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 16 to 112, higher (positive) score more severe pathology. Data show change from baseline to week 4.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
Units on a scale | -2.1 (0.49) | -2.2 (0.50) | -1.4 (0.48) | -2.8 (0.49)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2664, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3528, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0380, ANCOVA

32. Secondary Outcome: Mean Change From Baseline to Week 8 on the Positive and Negative Syndrome Scale (PANSS) General Psychopathology Scale Score
Description: PANSS rates psychopathology severity in schizophrenics. 16 items form a General Psychopathology scale:somatic concern, anxiety, guilt feeling, tension, mannerisms/posturing, depression, motor retardation, uncooperative, unusual thoughts, disorientation, poor attention, poor judgment/insight, disturbance of volition, poor impulse control, preoccupation, social avoidance. Scored on severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 16 to 112, higher (positive) score more severe pathology. Data show change from baseline to week 8.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
Units on a scale | -2.2 (0.52) | -2.3 (0.52) | -1.7 (0.50) | -2.9 (0.51)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3316, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3490, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0926, ANCOVA

33. Secondary Outcome: Mean Change From Baseline to Week 12 on the Positive and Negative Syndrome Scale (PANSS) General Psychopathology Scale Score
Description: PANSS rates psychopathology severity in schizophrenics. 16 items form a General Psychopathology scale:somatic concern, anxiety, guilt feeling, tension, mannerisms/posturing, depression, motor retardation, uncooperative, unusual thoughts, disorientation, poor attention, poor judgment/insight, disturbance of volition, poor impulse control, preoccupation, social avoidance. Scored on severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 16 to 112, higher (positive) score more severe pathology. Data show change from baseline to week 12.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Units on a scale | -2.4 (0.60) | -2.5 (0.61) | -1.1 (0.59) | -2.6 (0.60)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8835, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9748, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0883, ANCOVA

34. Secondary Outcome: Mean Change From Baseline to Week 16 on the Positive and Negative Syndrome Scale (PANSS) General Psychopathology Scale Score
Description: PANSS rates psychopathology severity in schizophrenics. 16 items form a General Psychopathology scale:somatic concern, anxiety, guilt feeling, tension, mannerisms/posturing, depression, motor retardation, uncooperative, unusual thoughts, disorientation, poor attention, poor judgment/insight, disturbance of volition, poor impulse control, preoccupation, social avoidance. Scored on severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 16 to 112, higher (positive) score more severe pathology. Data show change from baseline to week 16.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
Units on a scale | -2.6 (0.62) | -2.1 (0.67) | -1.9 (0.63) | -3.0 (0.63)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6948, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3345, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2447, ANCOVA

35. Secondary Outcome: Mean Change From Baseline to Week 20 on the Positive and Negative Syndrome Scale (PANSS) General Psychopathology Scale Score
Description: PANSS rates psychopathology severity in schizophrenics. 16 items form a General Psychopathology scale:somatic concern, anxiety, guilt feeling, tension, mannerisms/posturing, depression, motor retardation, uncooperative, unusual thoughts, disorientation, poor attention, poor judgment/insight, disturbance of volition, poor impulse control, preoccupation, social avoidance. Scored on severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 16 to 112, higher (positive) score more severe pathology. Data show change from baseline to week 20.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
Units on a scale | -2.9 (0.62) | -2.3 (0.67) | -2.3 (0.65) | -3.4 (0.63)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6115, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2233, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2343, ANCOVA

36. Secondary Outcome: Mean Change From Baseline to Week 24 on the Positive and Negative Syndrome Scale (PANSS) General Psychopathology Scale Score
Description: PANSS rates psychopathology severity in schizophrenics. 16 items form a General Psychopathology scale:somatic concern, anxiety, guilt feeling, tension, mannerisms/posturing, depression, motor retardation, uncooperative, unusual thoughts, disorientation, poor attention, poor judgment/insight, disturbance of volition, poor impulse control, preoccupation, social avoidance. Scored on severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 16 to 112, higher (positive) score more severe pathology. Data show change from baseline to week 24.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
Units on a scale | -3.0 (0.64) | -3.1 (0.69) | -2.3 (0.66) | -3.2 (0.64)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8228, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9373, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3190, ANCOVA

37. Secondary Outcome: Mean Change From Baseline to Endpoint From Negative Symptom Dimension Scores From the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates the severity of psychopathology in patients with schizophrenia. The negative symptoms factor score includes 5 negative symptoms (blunted affect, emotional withdrawal, poor rapport, positive/apathetic social withdrawal, lack of spontaneity) and 2 general psychopathology symptoms (motor retardation, active social avoidance). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 7 to 49. Higher (positive) score indicates worsening. Data represents change from baseline to endpoint.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
Units on a scale | -2.2 (0.43) | -2.1 (0.44) | -2.4 (0.43) | -2.2 (0.43)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9769, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8374, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7061, ANCOVA

38. Secondary Outcome: Mean Change From Baseline to Week 1 of Negative Symptom Dimension Scores From the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates the severity of psychopathology in patients with schizophrenia. The negative symptoms factor score includes 5 negative symptoms (blunted affect, emotional withdrawal, poor rapport, positive/apathetic social withdrawal, lack of spontaneity) and 2 general psychopathology symptoms (motor retardation, active social avoidance). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 7 to 49. Higher (positive) score indicates worsening. Data represents change from baseline to week 1.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
Units on a scale | -1.3 (0.28) | -1.0 (0.28) | -0.9 (0.28) | -1.3 (0.28)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9577, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5106, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2655, ANCOVA

39. Secondary Outcome: Mean Change From Baseline to Week 2 of Negative Symptom Dimension Scores From the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates the severity of psychopathology in patients with schizophrenia. The negative symptoms factor score includes 5 negative symptoms (blunted affect, emotional withdrawal, poor rapport, positive/apathetic social withdrawal, lack of spontaneity) and 2 general psychopathology symptoms (motor retardation, active social avoidance). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 7 to 49. Higher (positive) score indicates worsening. Data represents change from baseline to week 2.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
Units on a scale | -1.7 (0.33) | -1.5 (0.34) | -1.3 (0.33) | -2.1 (0.33)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3825, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2003, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0625, ANCOVA

40. Secondary Outcome: Mean Change From Baseline to Week 4 of Negative Symptom Dimension Scores From the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates the severity of psychopathology in patients with schizophrenia. The negative symptoms factor score includes 5 negative symptoms (blunted affect, emotional withdrawal, poor rapport, positive/apathetic social withdrawal, lack of spontaneity) and 2 general psychopathology symptoms (motor retardation, active social avoidance). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 7 to 49. Higher (positive) score indicates worsening. Data represents change from baseline to week 4.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
Units on a scale | -2.5 (0.39) | -1.6 (0.40) | -1.7 (0.38) | -3.0 (0.39)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2981, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0104, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0150, ANCOVA

41. Secondary Outcome: Mean Change From Baseline to Week 8 of Negative Symptom Dimension Scores From the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates the severity of psychopathology in patients with schizophrenia. The negative symptoms factor score includes 5 negative symptoms (blunted affect, emotional withdrawal, poor rapport, positive/apathetic social withdrawal, lack of spontaneity) and 2 general psychopathology symptoms (motor retardation, active social avoidance). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 7 to 49. Higher (positive) score indicates worsening. Data represents change from baseline to week 8.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
Units on a scale | -2.6 (0.44) | -1.9 (0.45) | -2.4 (0.43) | -3.0 (0.44)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4608, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0807, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2959, ANCOVA

42. Secondary Outcome: Mean Change From Baseline to Week 12 of Negative Symptom Dimension Scores From the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates the severity of psychopathology in patients with schizophrenia. The negative symptoms factor score includes 5 negative symptoms (blunted affect, emotional withdrawal, poor rapport, positive/apathetic social withdrawal, lack of spontaneity) and 2 general psychopathology symptoms (motor retardation, active social avoidance). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 7 to 49. Higher (positive) score indicates worsening. Data represents change from baseline to week 12.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Units on a scale | -2.8 (0.46) | -1.8 (0.47) | -2.6 (0.46) | -2.5 (0.46)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6759, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2418, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9808, ANCOVA

43. Secondary Outcome: Mean Change From Baseline to Week 16 of Negative Symptom Dimension Scores From the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates the severity of psychopathology in patients with schizophrenia. The negative symptoms factor score includes 5 negative symptoms (blunted affect, emotional withdrawal, poor rapport, positive/apathetic social withdrawal, lack of spontaneity) and 2 general psychopathology symptoms (motor retardation, active social avoidance). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 7 to 49. Higher (positive) score indicates worsening. Data represents change from baseline to week 16.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
Units on a scale | -3.2 (0.48) | -2.4 (0.52) | -2.6 (0.49) | -3.0 (0.49)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7599, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4543, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6040, ANCOVA

44. Secondary Outcome: Mean Change From Baseline to Week 20 of Negative Symptom Dimension Scores From the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates the severity of psychopathology in patients with schizophrenia. The negative symptoms factor score includes 5 negative symptoms (blunted affect, emotional withdrawal, poor rapport, positive/apathetic social withdrawal, lack of spontaneity) and 2 general psychopathology symptoms (motor retardation, active social avoidance). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 7 to 49. Higher (positive) score indicates worsening. Data represents change from baseline to week 20.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
Units on a scale | -3.6 (0.49) | -2.8 (0.53) | -2.8 (0.52) | -2.7 (0.50)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2476, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9490, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9035, ANCOVA

45. Secondary Outcome: Mean Change From Baseline to Week 24 of Negative Symptom Dimension Scores From the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates the severity of psychopathology in patients with schizophrenia. The negative symptoms factor score includes 5 negative symptoms (blunted affect, emotional withdrawal, poor rapport, positive/apathetic social withdrawal, lack of spontaneity) and 2 general psychopathology symptoms (motor retardation, active social avoidance). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 7 to 49. Higher (positive) score indicates worsening. Data represents change from baseline to week 24.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
Units on a scale | -2.7 (0.54) | -2.6 (0.58) | -2.3 (0.55) | -2.7 (0.54)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9472, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8335, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5674, ANCOVA

46. Secondary Outcome: Mean Change From Baseline to Endpoint of Positive Symptom Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in patients with schizophrenia. The positive symptoms dimension is the sum of 4 positive symptoms (delusions, hallucinatory behavior, grandiosity, suspiciousness/persecution), 1 negative symptom (stereotyped thinking), and 3 general psychopathology symptoms (somatic concern, unusual thought content, lack of judgment/insight). Each item scored on 7-point scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 8 to 56. Higher (positive) scores indicate worsening. Data show change from baseline to endpoint.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
Units on a scale | -0.3 (0.46) | -0.5 (0.47) | -0.5 (0.46) | 0.3 (0.46)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3536, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1940, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2129, ANCOVA

47. Secondary Outcome: Mean Change From Baseline to Week 1 of Positive Symptom Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in patients with schizophrenia. Positive symptoms dimension is the sum of 4 positive symptoms (delusions, hallucinatory behavior, grandiosity, suspiciousness/persecution), 1 negative symptom (stereotyped thinking), and 3 general psychopathology symptoms (somatic concern, unusual thought content, lack of judgment/insight). Each item is scored on a 7-point scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 8 to 56. Higher (positive) scores indicate worsening. Data show change from baseline to week 1.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
Units on a scale | -0.3 (0.25) | -0.6 (0.26) | 0.1 (0.25) | -0.5 (0.25)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5840, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6028, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1426, ANCOVA

48. Secondary Outcome: Mean Change From Baseline to Week 2 of Positive Symptom Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in patients with schizophrenia. The positive symptoms dimension is sum of 4 positive symptoms (delusions, hallucinatory behavior, grandiosity, suspiciousness/persecution), 1 negative symptom (stereotyped thinking), and 3 general psychopathology symptoms (somatic concern, unusual thought content, lack of judgment/insight). Each item is scored on a 7-point scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 8 to 56. Higher (positive) scores indicate worsening. Data show change from baseline to week 2.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
Units on a scale | -1.0 (0.30) | -0.9 (0.31) | -0.2 (0.29) | -0.8 (0.30)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5989, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7411, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1566, ANCOVA

49. Secondary Outcome: Mean Change From Baseline to Week 4 of Positive Symptom Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in patients with schizophrenia. The positive symptoms dimension is sum of 4 positive symptoms (delusions, hallucinatory behavior, grandiosity, suspiciousness/persecution), 1 negative symptom (stereotyped thinking), and 3 general psychopathology symptoms (somatic concern, unusual thought content, lack of judgment/insight). Each item is scored on a 7-point scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 8 to 56. Higher (positive) scores indicate worsening. Data show change from baseline to week 4.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
Units on a scale | -0.9 (0.31) | -1.0 (0.32) | -0.7 (0.30) | -1.3 (0.31)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2610, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4457, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1342, ANCOVA

50. Secondary Outcome: Mean Change From Baseline to Week 8 of Positive Symptom Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in patients with schizophrenia. The positive symptoms dimension is sum of 4 positive symptoms (delusions, hallucinatory behavior, grandiosity, suspiciousness/persecution), 1 negative symptom (stereotyped thinking), and 3 general psychopathology symptoms (somatic concern, unusual thought content, lack of judgment/insight). Each item is scored on a 7-point scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 8 to 56. Higher (positive) scores indicate worsening. Data show change from baseline to week 8.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
Units on a scale | -0.8 (0.35) | -1.4 (0.35) | -0.9 (0.33) | -1.6 (0.34)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0974, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6640, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1507, ANCOVA

51. Secondary Outcome: Mean Change From Baseline to Week 12 of Positive Symptom Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in patients with schizophrenia. The positive symptoms dimension is sum of 4 positive symptoms (delusions, hallucinatory behavior, grandiosity, suspiciousness/persecution), 1 negative symptom (stereotyped thinking), and 3 general psychopathology symptoms (somatic concern, unusual thought content, lack of judgment/insight). Each item is scored on a 7-point scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 8 to 56. Higher (positive) scores indicate worsening. Data show change from baseline to week 12.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Units on a scale | -0.9 (0.37) | -1.4 (0.38) | -0.7 (0.37) | -1.0 (0.38)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7649, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4866, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5002, ANCOVA

52. Secondary Outcome: Mean Change From Baseline to Week 16 of Positive Symptom Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in patients with schizophrenia. The positive symptoms dimension is sum of 4 positive symptoms (delusions, hallucinatory behavior, grandiosity, suspiciousness/persecution), 1 negative symptom (stereotyped thinking), and 3 general psychopathology symptoms (somatic concern, unusual thought content, lack of judgment/insight). Each item is scored on a 7-point scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 8 to 56. Higher (positive) scores indicate worsening. Data show change from baseline to week 16.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
Units on a scale | -0.9 (0.39) | -1.6 (0.42) | -0.9 (0.40) | -1.6 (0.40)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2076, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9355, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1890, ANCOVA

53. Secondary Outcome: Mean Change From Baseline to Week 20 of Positive Symptom Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in patients with schizophrenia. The positive symptoms dimension is sum of 4 positive symptoms (delusions, hallucinatory behavior, grandiosity, suspiciousness/persecution), 1 negative symptom (stereotyped thinking), and 3 general psychopathology symptoms (somatic concern, unusual thought content, lack of judgment/insight). Each item is scored on a 7-point scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 8 to 56. Higher (positive) scores indicate worsening. Data show change from baseline to week 20.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
Units on a scale | -1.4 (0.40) | -1.8 (0.44) | -1.2 (0.42) | -1.7 (0.41)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6320, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8777, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4378, ANCOVA

54. Secondary Outcome: Mean Change From Baseline to Week 24 of Positive Symptom Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in patients with schizophrenia. The positive symptoms dimension is sum of 4 positive symptoms (delusions, hallucinatory behavior, grandiosity, suspiciousness/persecution), 1 negative symptom (stereotyped thinking), and 3 general psychopathology symptoms (somatic concern, unusual thought content, lack of judgment/insight). Each item is scored on a 7-point scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 8 to 56. Higher (positive) scores indicate worsening. Data show change from baseline to week 24.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
Units on a scale | -1.0 (0.45) | -1.8 (0.49) | -0.8 (0.46) | -1.3 (0.45)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5544, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4446, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4483, ANCOVA

55. Secondary Outcome: Mean Change From Baseline to Endpoint From Anxiety/Depression Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The anxiety/depression dimension is the sum of 4 general psychopathology symptoms (anxiety, guilt feelings, tension, depression). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to endpoint. Higher (positive) scores indicate worsening.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
Units on a scale | -0.6 (0.30) | -0.5 (0.30) | -0.0 (0.29) | -0.0 (0.30)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1914, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2543, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9748, ANCOVA

56. Secondary Outcome: Mean Change From Baseline to Week 1 From Anxiety/Depression Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The anxiety/depression dimension is the sum of 4 general psychopathology symptoms (anxiety, guilt feelings, tension, depression). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 1. Higher (positive) scores indicate worsening.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
Units on a scale | -0.2 (0.21) | -0.3 (0.22) | -0.1 (0.21) | -0.4 (0.21)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5312, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7522, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3183, ANCOVA

57. Secondary Outcome: Mean Change From Baseline to Week 2 From Anxiety/Depression Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The anxiety/depression dimension is the sum of 4 general psychopathology symptoms (anxiety, guilt feelings, tension, depression). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 2. Higher (positive) scores indicate worsening.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
Units on a scale | -0.9 (0.22) | -0.7 (0.22) | -0.3 (0.21) | -0.7 (0.22)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5879, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8910, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1795, ANCOVA

58. Secondary Outcome: Mean Change From Baseline to Week 4 From Anxiety/Depression Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The anxiety/depression dimension is the sum of 4 general psychopathology symptoms (anxiety, guilt feelings, tension, depression). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 4. Higher (positive) scores indicate worsening.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
Units on a scale | -0.6 (0.26) | -0.8 (0.26) | -0.5 (0.25) | -0.7 (0.26)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6378, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8679, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5489, ANCOVA

59. Secondary Outcome: Mean Change From Baseline to Week 8 From Anxiety/Depression Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The anxiety/depression dimension is the sum of 4 general psychopathology symptoms (anxiety, guilt feelings, tension, depression). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 8. Higher (positive) scores indicate worsening.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
Units on a scale | -0.6 (0.27) | -0.6 (0.27) | -0.4 (0.26) | -0.6 (0.26)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9337, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9428, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5895, ANCOVA

60. Secondary Outcome: Mean Change From Baseline to Week 12 From Anxiety/Depression Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The anxiety/depression dimension is the sum of 4 general psychopathology symptoms (anxiety, guilt feelings, tension, depression). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 12. Higher (positive) scores indicate worsening.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Units on a scale | -0.6 (0.31) | -0.5 (0.32) | -0.2 (0.30) | -0.7 (0.31)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8695, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6637, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3152, ANCOVA

61. Secondary Outcome: Mean Change From Baseline to Week 16 From Anxiety/Depression Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The anxiety/depression dimension is the sum of 4 general psychopathology symptoms (anxiety, guilt feelings, tension, depression). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 16. Higher (positive) scores indicate worsening.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
Units on a scale | -0.6 (0.30) | -0.8 (0.32) | -0.9 (0.30) | -0.5 (0.30)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7472, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4503, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3127, ANCOVA

62. Secondary Outcome: Mean Change From Baseline to Week 20 From Anxiety/Depression Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The anxiety/depression dimension is the sum of 4 general psychopathology symptoms (anxiety, guilt feelings, tension, depression). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 20. Higher (positive) scores indicate worsening.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
Units on a scale | -0.6 (0.32) | -0.3 (0.34) | -0.4 (0.33) | -0.7 (0.32)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9193, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4814, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6097, ANCOVA

63. Secondary Outcome: Mean Change From Baseline to Week 24 From Anxiety/Depression Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The anxiety/depression dimension is the sum of 4 general psychopathology symptoms (anxiety, guilt feelings, tension, depression). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 24. Higher (positive) scores indicate worsening.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
Units on a scale | -0.9 (0.32) | -1.0 (0.35) | -0.5 (0.33) | -0.8 (0.32)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8594, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6157, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4846, ANCOVA

64. Secondary Outcome: Mean Change From Baseline to Endpoint From Disorganized Thought Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in schizophrenic patients. Disorganized thought dimension is the sum of 1 positive symptom (conceptual disorganization), 1 negative symptom (difficulty in abstract thinking), and 5 general psychopathology symptoms (mannerisms/posturing, disorientation, poor attention, disturbance of volition, preoccupation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 7 to 49. Higher (positive) score indicates worsening. Data indicates change from baseline to endpoint.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
Units on a scale | -0.3 (0.33) | -0.8 (0.33) | -0.7 (0.33) | -0.6 (0.33)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6076, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5827, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7865, ANCOVA

65. Secondary Outcome: Mean Change From Baseline to Week 1 From Disorganized Thought Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in schizophrenics. Disorganized thought dimension is the sum of 1 positive symptom (conceptual disorganization), 1 negative symptom (difficulty in abstract thinking), and 5 general psychopathology symptoms (mannerisms and posturing, disorientation, poor attention, disturbance of volition, preoccupation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 7 to 49. Higher (positive) score indicates worsening. Data indicates change from baseline to week 1.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
Units on a scale | -0.4 (0.22) | -0.1 (0.22) | -0.1 (0.21) | -0.7 (0.21)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3045, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0617, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0580, ANCOVA

66. Secondary Outcome: Mean Change From Baseline to Week 2 From Disorganized Thought Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in schizophrenics. Disorganized thought dimension is the sum of 1 positive symptom (conceptual disorganization), 1 negative symptom (difficulty in abstract thinking), and 5 general psychopathology symptoms (mannerisms and posturing, disorientation, poor attention, disturbance of volition, preoccupation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 7 to 49. Higher (positive) score indicates worsening. Data indicates change from baseline to week 2.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
Units on a scale | -0.2 (0.24) | -0.5 (0.24) | -0.4 (0.23) | -0.9 (0.24)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0194, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2270, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1181, ANCOVA

67. Secondary Outcome: Mean Change From Baseline to Week 4 From Disorganized Thought Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in schizophrenics. Disorganized thought dimension is the sum of 1 positive symptom (conceptual disorganization), 1 negative symptom (difficulty in abstract thinking), and 5 general psychopathology symptoms (mannerisms and posturing, disorientation, poor attention, disturbance of volition, preoccupation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 7 to 49. Higher (positive) score indicates worsening. Data indicates change from baseline to week 4.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
Units on a scale | -0.8 (0.24) | -0.6 (0.25) | -0.5 (0.24) | -1.3 (0.24)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1348, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0419, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0146, ANCOVA

68. Secondary Outcome: Mean Change From Baseline to Week 8 From Disorganized Thought Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in schizophrenics. Disorganized thought dimension is the sum of 1 positive symptom (conceptual disorganization), 1 negative symptom (difficulty in abstract thinking), and 5 general psychopathology symptoms (mannerisms and posturing, disorientation, poor attention, disturbance of volition, preoccupation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 7 to 49. Higher (positive) score indicates worsening. Data indicates change from baseline to week 8.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
Units on a scale | -0.7 (0.29) | -1.0 (0.29) | -0.7 (0.28) | -1.3 (0.28)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1292, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3773, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1348, ANCOVA

69. Secondary Outcome: Mean Change From Baseline to Week 12 From Disorganized Thought Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in schizophrenics. Disorganized thought dimension is the sum of 1 positive symptom (conceptual disorganization), 1 negative symptom (difficulty in abstract thinking), and 5 general psychopathology symptoms (mannerisms and posturing, disorientation, poor attention, disturbance of volition, preoccupation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 7 to 49. Higher (positive) score indicates worsening. Data indicates change from baseline to week 12.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Units on a scale | -1.2 (0.32) | -1.4 (0.33) | -0.6 (0.32) | -1.2 (0.32)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9642, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7814, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1455, ANCOVA

70. Secondary Outcome: Mean Change From Baseline to Week 16 From Disorganized Thought Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in schizophrenics. Disorganized thought dimension is the sum of 1 positive symptom (conceptual disorganization), 1 negative symptom (difficulty in abstract thinking), and 5 general psychopathology symptoms (mannerisms and posturing, disorientation, poor attention, disturbance of volition, preoccupation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 7 to 49. Higher (positive) score indicates worsening. Data indicates change from baseline to week 16.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
Units on a scale | -1.3 (0.33) | -0.8 (0.35) | -0.6 (0.33) | -1.5 (0.33)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5722, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1352, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0630, ANCOVA

71. Secondary Outcome: Mean Change From Baseline to Week 20 From Disorganized Thought Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in schizophrenics. Disorganized thought dimension is the sum of 1 positive symptom (conceptual disorganization), 1 negative symptom (difficulty in abstract thinking), and 5 general psychopathology symptoms (mannerisms and posturing, disorientation, poor attention, disturbance of volition, preoccupation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 7 to 49. Higher (positive) score indicates worsening. Data indicates change from baseline to week 20.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
Units on a scale | -1.3 (0.34) | -1.1 (0.37) | -1.2 (0.36) | -1.7 (0.35)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4607, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2538, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3406, ANCOVA

72. Secondary Outcome: Mean Change From Baseline to Week 24 From Disorganized Thought Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS rates severity of psychopathology in schizophrenics. Disorganized thought dimension is the sum of 1 positive symptom (conceptual disorganization), 1 negative symptom (difficulty in abstract thinking), and 5 general psychopathology symptoms (mannerisms and posturing, disorientation, poor attention, disturbance of volition, preoccupation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores range from 7 to 49. Higher (positive) score indicates worsening. Data indicates change from baseline to week 24.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
Units on a scale | -1.3 (0.34) | -1.2 (0.37) | -1.3 (0.35) | -1.4 (0.34)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8116, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6870, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8112, ANCOVA

73. Secondary Outcome: Mean Change From Baseline to Endpoint From the Hostility/Excitement Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The hostility/excitement dimension is the sum of 2 positive symptoms (excitement, hostility) and 2 general psychopathology symptoms (uncooperativeness, poor impulse control). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to endpoint. Higher (positive) score indicates worsening.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
Units on a scale | 0.0 (0.25) | 0.2 (0.25) | 0.3 (0.25) | 0.0 (0.25)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9786, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5879, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3973, ANCOVA

74. Secondary Outcome: Mean Change From Baseline to Week 1 From the Hostility/Excitement Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The hostility/excitement dimension is the sum of 2 positive symptoms (excitement, hostility) and 2 general psychopathology symptoms (uncooperativeness, poor impulse control). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 1. Higher (positive) score indicates worsening.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
Units on a scale | 0.1 (0.16) | -0.3 (0.17) | 0.0 (0.16) | -0.1 (0.16)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4030, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3777, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6493, ANCOVA

75. Secondary Outcome: Mean Change From Baseline to Week 2 From the Hostility/Excitement Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The hostility/excitement dimension is the sum of 2 positive symptoms (excitement, hostility) and 2 general psychopathology symptoms (uncooperativeness, poor impulse control). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 2. Higher (positive) score indicates worsening.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
Units on a scale | -0.3 (0.19) | -0.2 (0.19) | 0.2 (0.19) | -0.3 (0.19)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9871, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5859, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0328, ANCOVA

76. Secondary Outcome: Mean Change From Baseline to Week 4 From the Hostility/Excitement Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The hostility/excitement dimension is the sum of 2 positive symptoms (excitement, hostility) and 2 general psychopathology symptoms (uncooperativeness, poor impulse control). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 4. Higher (positive) score indicates worsening.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
Units on a scale | -0.1 (0.16) | -0.5 (0.17) | -0.2 (0.16) | -0.4 (0.16)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2318, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6211, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3125, ANCOVA

77. Secondary Outcome: Mean Change From Baseline to Week 8 From the Hostility/Excitement Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The hostility/excitement dimension is the sum of 2 positive symptoms (excitement, hostility) and 2 general psychopathology symptoms (uncooperativeness, poor impulse control). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 8. Higher (positive) score indicates worsening.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
Units on a scale | -0.1 (0.20) | -0.3 (0.20) | -0.3 (0.19) | -0.5 (0.20)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2425, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6597, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4753, ANCOVA

78. Secondary Outcome: Mean Change From Baseline to Week 12 From the Hostility/Excitement Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The hostility/excitement dimension is the sum of 2 positive symptoms (excitement, hostility) and 2 general psychopathology symptoms (uncooperativeness, poor impulse control). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 12. Higher (positive) score indicates worsening.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Units on a scale | -0.1 (0.22) | -0.2 (0.23) | 0.3 (0.22) | -0.5 (0.22)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1715, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3056, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0083, ANCOVA

79. Secondary Outcome: Mean Change From Baseline to Week 16 From the Hostility/Excitement Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The hostility/excitement dimension is the sum of 2 positive symptoms (excitement, hostility) and 2 general psychopathology symptoms (uncooperativeness, poor impulse control). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 16. Higher (positive) score indicates worsening.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
Units on a scale | -0.1 (0.23) | 0.1 (0.25) | 0.2 (0.24) | -0.4 (0.24)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2681, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1475, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0647, ANCOVA

80. Secondary Outcome: Mean Change From Baseline to Week 20 From the Hostility/Excitement Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The hostility/excitement dimension is the sum of 2 positive symptoms (excitement, hostility) and 2 general psychopathology symptoms (uncooperativeness, poor impulse control). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 20. Higher (positive) score indicates worsening.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
Units on a scale | -0.1 (0.21) | -0.1 (0.23) | -0.3 (0.22) | -0.5 (0.22)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1670, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1737, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3720, ANCOVA

81. Secondary Outcome: Mean Change From Baseline to Week 24 From the Hostility/Excitement Dimension of the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. The hostility/excitement dimension is the sum of 2 positive symptoms (excitement, hostility) and 2 general psychopathology symptoms (uncooperativeness, poor impulse control). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores may range from 4 to 28. The data presented here represents the change from baseline to week 24. Higher (positive) score indicates worsening.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
Units on a scale | -0.2 (0.24) | -0.4 (0.25) | 0.1 (0.24) | -0.5 (0.24)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3547, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6043, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0463, ANCOVA

82. Secondary Outcome: Change From Baseline to Endpoint in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to endpoint in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 68 | 71 | 70
Units on a scale | -0.1 (0.06) | -0.1 (0.06) | -0.2 (0.06) | -0.2 (0.06)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9258, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9116, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4848, ANCOVA

83. Secondary Outcome: Change From Baseline to Week 1 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 1 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
Units on a scale | -0.1 (0.03) | -0.1 (0.03) | -0.0 (0.03) | -0.1 (0.03)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7612, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5761, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1576, ANCOVA

84. Secondary Outcome: Change From Baseline to Week 2 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 2 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
Units on a scale | -0.1 (0.04) | -0.2 (0.04) | -0.1 (0.04) | -0.1 (0.04)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9565, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9178, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1491, ANCOVA

85. Secondary Outcome: Change From Baseline to Week 4 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 4 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
units on a scale | -0.2 (0.05) | -0.1 (0.05) | -0.1 (0.05) | -0.2 (0.05)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7056, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5179, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4585, ANCOVA

86. Secondary Outcome: Change From Baseline to Week 6 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 6 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 6
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 57 | 55 | 60 | 59
units on a scale | -0.1 (0.05) | -0.2 (0.05) | -0.1 (0.05) | -0.2 (0.05)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0690, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5324, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0946, ANCOVA

87. Secondary Outcome: Change From Baseline to Week 8 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 8 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
units on a scale | -0.1 (0.06) | -0.2 (0.06) | -0.2 (0.05) | -0.2 (0.05)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1878, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4294, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6504, ANCOVA

88. Secondary Outcome: Change From Baseline to Week 10 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 10 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 10
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 50 | 56 | 53
units on a scale | -0.2 (0.06) | -0.2 (0.06) | -0.2 (0.06) | -0.3 (0.06)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4022, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6246, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8655, ANCOVA

89. Secondary Outcome: Change From Baseline to Week 12 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 12 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
units on a scale | -0.2 (0.06) | -0.2 (0.06) | -0.3 (0.06) | -0.2 (0.06)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5676, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5239, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4092, ANCOVA

90. Secondary Outcome: Change From Baseline to Week 14 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 14 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 14
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 47 | 52 | 50
units on a scale | -0.2 (0.06) | -0.2 (0.06) | -0.3 (0.06) | -0.3 (0.06)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5195, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1732, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7455, ANCOVA

91. Secondary Outcome: Change From Baseline to Week 16 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 16 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
units on a scale | -0.2 (0.06) | -0.2 (0.07) | -0.3 (0.06) | -0.3 (0.06)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6885, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5443, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9343, ANCOVA

92. Secondary Outcome: Change From Baseline to Week 18 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 18 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 18
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 42 | 47 | 49
units on a scale | -0.3 (0.06) | -0.2 (0.07) | -0.3 (0.06) | -0.3 (0.06)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9093, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4701, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9764, ANCOVA

93. Secondary Outcome: Change From Baseline to Week 20 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 20 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
units on a scale | -0.2 (0.06) | -0.2 (0.07) | -0.3 (0.07) | -0.3 (0.07)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8115, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5378, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9144, ANCOVA

94. Secondary Outcome: Change From Baseline to Week 22 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 22 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 22
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 47 | 41 | 44 | 46
units on a scale | -0.3 (0.07) | -0.2 (0.07) | -0.3 (0.07) | -0.3 (0.07)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9812, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5464, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8811, ANCOVA

95. Secondary Outcome: Change From Baseline to Week 24 in the Clinical Global Impression of Severity of Illness (CGI-S) Rating
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness. The data presented represents the change from baseline to week 24 in the CGI-S rating. A negative value indicates improvement.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 45
units on a scale | -0.3 (0.07) | -0.2 (0.07) | -0.3 (0.07) | -0.3 (0.07)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6487, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4204, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6955, ANCOVA

96. Secondary Outcome: Mean Change From Baseline to Endpoint in Personal and Social Performance Scale (PSP) Scores
Description: PSP is a validated clinician-rated assessment of functioning. Four areas of functioning (socially useful activities, personal/social relationships, self-care, disturbing/aggressive behaviors) are assessed on a 6-point scale (0=absent to 5=very severe). A transformed score from 1 to 100 is generated from the raw score based on the clinical interpretation of the scores generated in the 4 areas of functioning, with a higher transformed score indicating better function. Data presented here represents change from baseline to endpoint in the overall score with positive values signifying improvement.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 66 | 64 | 67 | 66
units on a scale | 1.5 (0.98) | 2.1 (0.99) | 2.2 (0.97) | 2.2 (0.98)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6042, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9783, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9739, ANCOVA

97. Secondary Outcome: Mean Change From Baseline to Week 4 in Personal and Social Performance Scale (PSP) Scores
Description: PSP is a validated clinician-rated assessment of functioning. Four areas of functioning (socially useful activities, personal/social relationships, self-care, disturbing/aggressive behaviors) are assessed on a 6-point scale (0=absent to 5=very severe). A transformed score from 1 to 100 is generated from the raw score based on the clinical interpretation of the scores generated in the 4 areas of functioning, with a higher transformed score indicating better function. Data presented here represents change from baseline to week 4 in the overall score with positive values signifying improvement.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
units on a scale | 1.7 (0.65) | 2.4 (0.67) | 2.0 (0.64) | 2.5 (0.65)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3466, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8469, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5439, ANCOVA

98. Secondary Outcome: Mean Change From Baseline to Week 12 in Personal and Social Performance Scale (PSP) Scores
Description: PSP is a validated clinician-rated assessment of functioning. Four areas of functioning (socially useful activities, personal/social relationships, self-care, disturbing/aggressive behaviors) are assessed on a 6-point scale (0=absent to 5=very severe). A transformed score from 1 to 100 is generated from the raw score based on the clinical interpretation of the scores generated in the 4 areas of functioning, with a higher transformed score indicating better function. Data presented here represents change from baseline to week 12 in the overall score with positive values signifying improvement.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
units on a scale | 3.1 (0.83) | 2.9 (0.85) | 3.4 (0.82) | 2.5 (0.84)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6059, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7474, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4424, ANCOVA

99. Secondary Outcome: Mean Change From Baseline to Week 24 in Personal and Social Performance Scale (PSP) Scores
Description: PSP is a validated clinician-rated assessment of functioning. Four areas of functioning (socially useful activities, personal/social relationships, self-care, disturbing/aggressive behaviors) are assessed on a 6-point scale (0=absent to 5=very severe). A transformed score from 1 to 100 is generated from the raw score based on the clinical interpretation of the scores generated in the 4 areas of functioning, with a higher transformed score indicating better function. Data presented here represents change from baseline to week 24 in the overall score with positive values signifying improvement.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 45
units on a scale | 2.0 (1.14) | 3.5 (1.22) | 3.2 (1.17) | 3.1 (1.15)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4874, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8243, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9562, ANCOVA

100. Secondary Outcome: Mean Change From Baseline to Endpoint in CNSVitalSigns Cognitive Battery Scores - Verbal Memory Test
Description: CNSVitalSigns cognitive battery consists of 4 tests (Verbal Memory, Symbol-Digit Coding Test, Shifting Attention Test, Continuous Performance Test [CPT]). With Verbal Memory Test, patient asked to remember 15 words within a field of 15 distractors immediately and after twenty minute delay. Score is the sum of correct immediate "hits", correct immediate "passes", correct delayed "hits", and correct delayed "passes". Total score may range from 0 to 60, with a higher score indicating more correct responses. Data represents change from baseline to endpoint, with positive score showing improvement.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 58 | 59 | 57 | 59
units on a scale | -1.2 (0.97) | -3.0 (0.96) | -0.4 (0.98) | 0.0 (0.96)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3686, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0270, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7322, ANCOVA

101. Secondary Outcome: Mean Change From Baseline to Week 12 in CNSVitalSigns Cognitive Battery Scores - Verbal Memory Test
Description: CNSVitalSigns cognitive battery consists of 4 tests (Verbal Memory, Symbol-Digit Coding Test, Shifting Attention Test, Continuous Performance Test [CPT]). With Verbal Memory Test, patient asked to remember 15 words within a field of 15 distractors immediately and after twenty minute delay. Score is the sum of correct immediate "hits", correct immediate "passes", correct delayed "hits", and correct delayed "passes". Total score may range from 0 to 60, with a higher score indicating more correct responses. Data represents change from baseline to week 12, with positive score showing improvement.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 46 | 52 | 49
units on a scale | -1.3 (1.11) | -0.4 (1.14) | -1.4 (1.08) | -0.2 (1.11)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4646, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8783, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4213, ANCOVA

102. Secondary Outcome: Mean Change From Baseline to Week 24 in CNSVitalSigns Cognitive Battery Scores - Verbal Memory Test
Description: CNSVitalSigns cognitive battery consists of 4 tests (Verbal Memory, Symbol-Digit Coding Test, Shifting Attention Test, Continuous Performance Test [CPT]). With Verbal Memory Test, patient asked to remember 15 words within a field of 15 distractors immediately and after twenty minute delay. Score is the sum of correct immediate "hits", correct immediate "passes", correct delayed "hits", and correct delayed "passes". Total score may range from 0 to 60, with a higher score indicating more correct responses. Data represents change from baseline to week 24, with positive score showing improvement.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 39 | 44 | 44
units on a scale | -0.1 (1.03) | -2.9 (1.11) | -0.1 (1.05) | 0.5 (1.05)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6597, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0262, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6652, ANCOVA

103. Secondary Outcome: Mean Change From Baseline to Endpoint in CNSVitalSigns Cognitive Battery Scores - Symbol-digit Coding Test (SDCT)
Description: Symbol-digit coding test (SDCT) is one test in the CNSVitalSigns cognitive battery. SDCT assesses speed of processing. Subject is taught to link numbers to digits. The test consists of serial presentations of screens, each of which contains a bank of 8 symbols above and 8 empty boxes below. The subject types in the number that corresponds to the symbol highlighted. Scoring is the number of correct responses generated in 2 minutes. A higher score indicates greater processing speed. Data represents change from baseline to endpoint with positive values representing improvement.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Number of correct responses
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 58 | 59 | 57 | 59
Number of correct responses | -2.0 (2.28) | -4.2 (2.25) | 0.8 (2.29) | 1.1 (2.25)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3355, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0953, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9235, ANCOVA

104. Secondary Outcome: Mean Change From Baseline to Week 12 in CNSVitalSigns Cognitive Battery Scores - Symbol-digit Coding Test
Description: Symbol-digit coding test (SDCT) is one test in the CNSVitalSigns cognitive battery. SDCT assesses speed of processing. Subject is taught to link numbers to digits. The test consists of serial presentations of screens, each of which contains a bank of 8 symbols above and 8 empty boxes below. The subject types in the number that corresponds to the symbol highlighted. Scoring is the number of correct responses generated in 2 minutes. A higher score indicates greater processing speed. Data represents change from baseline to week 12 with positive values representing improvement.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Number of correct responses
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 46 | 52 | 49
Number of correct responses | -1.3 (1.53) | -1.8 (1.58) | -0.4 (1.49) | 0.5 (1.53)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4164, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3003, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6907, ANCOVA

105. Secondary Outcome: Mean Change From Baseline to Week 24 in CNSVitalSigns Cognitive Battery Scores - Symbol-digit Coding Test
Description: Symbol-digit coding test (SDCT) is one test in the CNSVitalSigns cognitive battery. SDCT assesses speed of processing. Subject is taught to link numbers to digits. The test consists of serial presentations of screens, each of which contains a bank of 8 symbols above and 8 empty boxes below. The subject types in the number that corresponds to the symbol highlighted. Scoring is the number of correct responses generated in 2 minutes. A higher score indicates greater processing speed. Data represents change from baseline to week 24 with positive values representing improvement.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Number of correct responses
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 39 | 43 | 44
Number of correct responses | -2.3 (2.85) | -5.2 (3.08) | 0.0 (2.94) | 2.4 (2.90)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2518, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0739, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5644, ANCOVA

106. Secondary Outcome: Mean Change From Baseline to Endpoint in CNSVitalSigns Cognitive Battery Scores - Shifting Attention Test
Description: The Shifting Attention Test is a test in the CNSVitalSigns cognitive battery. The Shifting Attention Test assesses attention and executive function. Patients were instructed to match geometric objects either by shape or by color. Composite Scoring presented here was calculated as the number of correct responses minus the number of errors. A higher score indicates more correct responses. The data represent the change from baseline to endpoint and a positive value represents improvement.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Correct responses minue errors
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 58 | 59 | 56 | 58
Correct responses minue errors | -3.1 (2.83) | 0.9 (2.79) | 1.5 (2.88) | 0.1 (2.81)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4305, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8299, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7283, ANCOVA

107. Secondary Outcome: Mean Change From Baseline to Week 12 in CNSVitalSigns Cognitive Battery Scores - Shifting Attention Test
Description: The Shifting Attention Test is a test in the CNSVitalSigns cognitive battery. The Shifting Attention Test assesses attention and executive function. Patients were instructed to match geometric objects either by shape or by color. Composite Scoring presented here was calculated as the number of correct responses minus the number of errors. A higher score indicates more correct responses. The data represent the change from baseline to week 12 and a positive value represents improvement.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Correct responses minus errors
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 48 | 46 | 51 | 48
Correct responses minus errors | 1.0 (2.32) | -1.7 (2.36) | 3.1 (2.25) | 0.0 (2.31)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7610, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6091, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3368, ANCOVA

108. Secondary Outcome: Mean Change From Baseline to Week 24 in CNSVitalSigns Cognitive Battery Scores - Shifting Attention Test
Description: The Shifting Attention Test is a test in the CNSVitalSigns cognitive battery. The Shifting Attention Test assesses attention and executive function. Patients were instructed to match geometric objects either by shape or by color. Composite Scoring presented here was calculated as the number of correct responses minus the number of errors. A higher score indicates more correct responses. The data represent the change from baseline to week 24 and a positive value represents improvement.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Correct responses minus errors
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 39 | 43 | 45
Correct responses minus errors | -1.8 (3.11) | 2.5 (3.34) | 0.9 (3.20) | -0.9 (3.11)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8457, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4531, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6867, ANCOVA

109. Secondary Outcome: Mean Change From Baseline to Endpoint in CNSVitalSigns Cognitive Battery Scores - 4-part Continuous Performance Test [CPT]
Description: The 4-Part Continuous Performance Test (CPT) is a component of the CNSVitalSigns cognitive battery. The 4-Part CPT assesses working memory. The patient was presented with targets and had to remember target presentation sequencing in order to respond to the directions. The complexity of the directions increased as the patient proceeded through the 4 parts of the test. Scoring is based on the number of correct responses, with a higher number indicating more correct responses. Data represents change from baseline to endpoint with positive values demonstrating improvement.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Correct responses
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 58 | 59 | 56 | 58
Correct responses | 0.0 (1.50) | -6.4 (1.49) | -1.3 (1.52) | 0.1 (1.50)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9705, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0021, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5013, ANCOVA

110. Secondary Outcome: Mean Change From Baseline to Week 12 in CNSVitalSigns Cognitive Battery Scores - 4-part Continuous Performance Test [CPT]
Description: The 4-Part Continuous Performance Test (CPT) is a component of the CNSVitalSigns cognitive battery. The 4-Part CPT assesses working memory. The patient was presented with targets and had to remember target presentation sequencing in order to respond to the directions. The complexity of the directions increased as the patient proceeded through the 4 parts of the test. Scoring is based on the number of correct responses, with a higher number indicating more correct responses. Data represents change from baseline to week 12 with positive values demonstrating improvement.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Correct responses
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 48 | 46 | 51 | 48
Correct responses | -0.3 (1.56) | -5.6 (1.59) | -3.1 (1.51) | 0.4 (1.55)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7330, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0068, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1040, ANCOVA

111. Secondary Outcome: Mean Change From Baseline to Week 24 in CNSVitalSigns Cognitive Battery Scores - 4-part Continuous Performance Test [CPT]
Description: The 4-Part Continuous Performance Test (CPT) is a component of the CNSVitalSigns cognitive battery. The 4-Part CPT assesses working memory. The patient was presented with targets and had to remember target presentation sequencing in order to respond to the directions. The complexity of the directions increased as the patient proceeded through the 4 parts of the test. Scoring is based on the number of correct responses, with a higher number indicating more correct responses. Data represents change from baseline to week 24 with positive values demonstrating improvement.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Least Squares Mean (Standard Error); unit: Correct responses
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 39 | 43 | 45
Correct responses | -0.2 (1.77) | -6.2 (1.92) | 0.5 (1.83) | 0.3 (1.79)
Statistical Analysis 1: Comparison: 150 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8220, ANCOVA
Statistical Analysis 2: Comparison: 200 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0144, ANCOVA
Statistical Analysis 3: Comparison: 250 mg/Day Armodafinil vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9464, ANCOVA

112. Secondary Outcome: Changes From Baseline to Endpoint in the Abnormal Involuntary Movement Scale (AIMS) Total Scores
Description: Abnormal Involuntary Movement Scale (AIMS) is a 14-item, clinician-rated scale to assess the severity of dyskinesias in patients taking neuroleptic drugs. Items 1 through 10 were rated using a 5-point (0-4) scale, items 11 through 14 were rated using a 2-point (no or yes) scale. The AIMS total score is the sum of items 1 through 10, and can range from 0-40. A higher score indicates a presence of more severe dyskinesias. Data represents change from baseline to endpoint, positive value represents worsening.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
units on a scale | 0.0 (1.15) | 0.0 (1.16) | 0.2 (1.44) | -0.2 (0.71)

113. Secondary Outcome: Changes From Baseline to Week 1 in the Abnormal Involuntary Movement Scale (AIMS) Total Scores
Description: Abnormal Involuntary Movement Scale (AIMS) is a 14-item, clinician-rated scale to assess the severity of dyskinesias in patients taking neuroleptic drugs. Items 1 through 10 were rated using a 5-point (0-4) scale, items 11 through 14 were rated using a 2-point (no or yes) scale. The AIMS total score is the sum of items 1 through 10, and can range from 0-40. A higher score indicates a presence of more severe dyskinesias. Data represents change from baseline to week 1, positive value represents worsening.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
units on a scale | -0.1 (0.46) | -0.1 (0.87) | 0.0 (0.69) | -0.1 (0.68)

114. Secondary Outcome: Changes From Baseline to Week 2 in the Abnormal Involuntary Movement Scale (AIMS) Total Scores
Description: Abnormal Involuntary Movement Scale (AIMS) is a 14-item, clinician-rated scale to assess the severity of dyskinesias in patients taking neuroleptic drugs. Items 1 through 10 were rated using a 5-point (0-4) scale, items 11 through 14 were rated using a 2-point (no or yes) scale. The AIMS total score is the sum of items 1 through 10, and can range from 0-40. A higher score indicates a presence of more severe dyskinesias. Data represents change from baseline to week 2, positive value represents worsening.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
units on a scale | -0.1 (0.48) | -0.1 (0.93) | 0.0 (0.70) | 0.0 (0.25)

115. Secondary Outcome: Changes From Baseline to Week 4 in the Abnormal Involuntary Movement Scale (AIMS) Total Scores
Description: Abnormal Involuntary Movement Scale (AIMS) is a 14-item, clinician-rated scale to assess the severity of dyskinesias in patients taking neuroleptic drugs. Items 1 through 10 were rated using a 5-point (0-4) scale, items 11 through 14 were rated using a 2-point (no or yes) scale. The AIMS total score is the sum of items 1 through 10, and can range from 0-40. A higher score indicates a presence of more severe dyskinesias. Data represents change from baseline to week 4, positive value represents worsening.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
units on a scale | 0.0 (0.71) | 0.0 (0.23) | -0.1 (0.53) | 0.0 (0.40)

116. Secondary Outcome: Changes From Baseline to Week 8 in the Abnormal Involuntary Movement Scale (AIMS) Total Scores
Description: Abnormal Involuntary Movement Scale (AIMS) is a 14-item, clinician-rated scale to assess the severity of dyskinesias in patients taking neuroleptic drugs. Items 1 through 10 were rated using a 5-point (0-4) scale, items 11 through 14 were rated using a 2-point (no or yes) scale. The AIMS total score is the sum of items 1 through 10, and can range from 0-40. A higher score indicates a presence of more severe dyskinesias. Data represents change from baseline to week 8, positive value represents worsening.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
units on a scale | 0.0 (0.75) | -0.1 (1.43) | 0.0 (0.76) | -0.1 (0.71)

117. Secondary Outcome: Changes From Baseline to Week 12 in the Abnormal Involuntary Movement Scale (AIMS) Total Scores
Description: Abnormal Involuntary Movement Scale (AIMS) is a 14-item, clinician-rated scale to assess the severity of dyskinesias in patients taking neuroleptic drugs. Items 1 through 10 were rated using a 5-point (0-4) scale, items 11 through 14 were rated using a 2-point (no or yes) scale. The AIMS total score is the sum of items 1 through 10, and can range from 0-40. A higher score indicates a presence of more severe dyskinesias. Data represents change from baseline to week 12, positive value represents worsening.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
units on a scale | 0.2 (1.06) | 0.0 (0.97) | 0.4 (2.31) | -0.1 (1.13)

118. Secondary Outcome: Changes From Baseline to Week 16 in the Abnormal Involuntary Movement Scale (AIMS) Total Scores
Description: Abnormal Involuntary Movement Scale (AIMS) is a 14-item, clinician-rated scale to assess the severity of dyskinesias in patients taking neuroleptic drugs. Items 1 through 10 were rated using a 5-point (0-4) scale, items 11 through 14 were rated using a 2-point (no or yes) scale. The AIMS total score is the sum of items 1 through 10, and can range from 0-40. A higher score indicates a presence of more severe dyskinesias. Data represents change from baseline to week 16, positive value represents worsening.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
units on a scale | 0.0 (0.88) | 0.2 (0.92) | 0.2 (1.25) | -0.3 (1.09)

119. Secondary Outcome: Changes From Baseline to Week 20 in the Abnormal Involuntary Movement Scale (AIMS) Total Scores
Description: Abnormal Involuntary Movement Scale (AIMS) is a 14-item, clinician-rated scale to assess the severity of dyskinesias in patients taking neuroleptic drugs. Items 1 through 10 were rated using a 5-point (0-4) scale, items 11 through 14 were rated using a 2-point (no or yes) scale. The AIMS total score is the sum of items 1 through 10, and can range from 0-40. A higher score indicates a presence of more severe dyskinesias. Data represents change from baseline to week 20, positive value represents worsening.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
units on a scale | -0.1 (0.95) | 0.3 (1.70) | 0.2 (1.53) | -0.3 (0.79)

120. Secondary Outcome: Changes From Baseline to Week 24 in the Abnormal Involuntary Movement Scale (AIMS) Total Scores
Description: Abnormal Involuntary Movement Scale (AIMS) is a 14-item, clinician-rated scale to assess the severity of dyskinesias in patients taking neuroleptic drugs. Items 1 through 10 were rated using a 5-point (0-4) scale, items 11 through 14 were rated using a 2-point (no or yes) scale. The AIMS total score is the sum of items 1 through 10, and can range from 0-40. A higher score indicates a presence of more severe dyskinesias. Data represents change from baseline to week 24, positive value represents worsening.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
units on a scale | -0.1 (1.10) | 0.1 (0.50) | 0.3 (1.75) | -0.2 (0.82)

121. Secondary Outcome: Changes From Baseline to Endpoint in the Simpson-Angus Extrapyramidal Symptoms (EPS) Scale Total Score
Description: The Simpson-Angus EPS Scale is a clinician-rated scale to assess parkinsonian and extrapyramidal symptoms (10 items) associated with antipsychotic medications. Each item is rated on a 5-point scale. In addition, this scale was used to evaluate and characterize adverse events of extrapyramidal symptoms. Total scores are calculated by summing the scores of each item (minimum 0, maximum 40) and dividing by the number of items (10). Scores can range from 0-4. A higher score indicates more severe symptoms. Data represents change from baseline to endpoint, positive values represent worsening.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
units on a scale | 0.0 (0.67) | 0.0 (0.61) | 0.2 (1.43) | -0.1 (0.62)

122. Secondary Outcome: Changes From Baseline to Week 1 in the Simpson-Angus Extrapyramidal Symptoms (EPS) Scale Total Score
Description: The Simpson-Angus EPS Scale is a clinician-rated scale to assess parkinsonian and extrapyramidal symptoms (10 items) associated with antipsychotic medications. Each item is rated on a 5-point scale. In addition, this scale was used to evaluate and characterize adverse events of extrapyramidal symptoms. Total scores are calculated by summing the scores of each item (minimum 0, maximum 40) and dividing by the number of items (10). Scores can range from 0-4. A higher score indicates more severe symptoms. Data represents change from baseline to week 1, positive values represent worsening.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
units on a scale | 0.0 (0.87) | -0.2 (0.6) | 0.1 (0.48) | 0.0 (0.54)

123. Secondary Outcome: Changes From Baseline to Week 2 in the Simpson-Angus Extrapyramidal Symptoms (EPS) Scale Total Score
Description: The Simpson-Angus EPS Scale is a clinician-rated scale to assess parkinsonian and extrapyramidal symptoms (10 items) associated with antipsychotic medications. Each item is rated on a 5-point scale. In addition, this scale was used to evaluate and characterize adverse events of extrapyramidal symptoms. Total scores are calculated by summing the scores of each item (minimum 0, maximum 40) and dividing by the number of items (10). Scores can range from 0-4. A higher score indicates more severe symptoms. Data represents change from baseline to week 2, positive values represent worsening.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
units on a scale | 0.0 (0.84) | -0.2 (0.54) | 0.0 (0.27) | -0.1 (0.52)

124. Secondary Outcome: Changes From Baseline to Week 4 in the Simpson-Angus Extrapyramidal Symptoms (EPS) Scale Total Score
Description: The Simpson-Angus EPS Scale is a clinician-rated scale to assess parkinsonian and extrapyramidal symptoms (10 items) associated with antipsychotic medications. Each item is rated on a 5-point scale. In addition, this scale was used to evaluate and characterize adverse events of extrapyramidal symptoms. Total scores are calculated by summing the scores of each item (minimum 0, maximum 40) and dividing by the number of items (10). Scores can range from 0-4. A higher score indicates more severe symptoms. Data represents change from baseline to week 4, positive values represent worsening.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
units on a scale | 0.0 (0.82) | -0.1 (0.53) | 0.0 (0.37) | 0.0 (0.38)

125. Secondary Outcome: Changes From Baseline to Week 8 in the Simpson-Angus Extrapyramidal Symptoms (EPS) Scale Total Score
Description: The Simpson-Angus EPS Scale is a clinician-rated scale to assess parkinsonian and extrapyramidal symptoms (10 items) associated with antipsychotic medications. Each item is rated on a 5-point scale. In addition, this scale was used to evaluate and characterize adverse events of extrapyramidal symptoms. Total scores are calculated by summing the scores of each item (minimum 0, maximum 40) and dividing by the number of items (10). Scores can range from 0-4. A higher score indicates more severe symptoms. Data represents change from baseline to week 8, positive values represent worsening.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
units on a scale | 0.1 (0.63) | -0.2 (0.97) | 0.1 (0.54) | -0.2 (0.58)

126. Secondary Outcome: Changes From Baseline to Week 12 in the Simpson-Angus Extrapyramidal Symptoms (EPS) Scale Total Score
Description: The Simpson-Angus EPS Scale is a clinician-rated scale to assess parkinsonian and extrapyramidal symptoms (10 items) associated with antipsychotic medications. Each item is rated on a 5-point scale. In addition, this scale was used to evaluate and characterize adverse events of extrapyramidal symptoms. Total scores are calculated by summing the scores of each item (minimum 0, maximum 40) and dividing by the number of items (10). Scores can range from 0-4. A higher score indicates more severe symptoms. Data represents change from baseline to week 12, positive values represent worsening.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
units on a scale | 0.1 (0.72) | -0.2 (1.02) | 0.1 (0.33) | -0.2 (0.67)

127. Secondary Outcome: Changes From Baseline to Week 16 in the Simpson-Angus Extrapyramidal Symptoms (EPS) Scale Total Score
Description: The Simpson-Angus EPS Scale is a clinician-rated scale to assess parkinsonian and extrapyramidal symptoms (10 items) associated with antipsychotic medications. Each item is rated on a 5-point scale. In addition, this scale was used to evaluate and characterize adverse events of extrapyramidal symptoms. Total scores are calculated by summing the scores of each item (minimum 0, maximum 40) and dividing by the number of items (10). Scores can range from 0-4. A higher score indicates more severe symptoms. Data represents change from baseline to week 16, positive values represent worsening.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
units on a scale | 0.0 (0.70) | -0.1 (0.53) | 0.0 (0.38) | -0.2 (0.66)

128. Secondary Outcome: Changes From Baseline to Week 20 in the Simpson-Angus Extrapyramidal Symptoms (EPS) Scale Total Score
Description: The Simpson-Angus EPS Scale is a clinician-rated scale to assess parkinsonian and extrapyramidal symptoms (10 items) associated with antipsychotic medications. Each item is rated on a 5-point scale. In addition, this scale was used to evaluate and characterize adverse events of extrapyramidal symptoms. Total scores are calculated by summing the scores of each item (minimum 0, maximum 40) and dividing by the number of items (10). Scores can range from 0-4. A higher score indicates more severe symptoms. Data represents change from baseline to week 20, positive values represent worsening.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
units on a scale | 0.0 (0.54) | -0.1 (0.51) | -0.1 (0.47) | -0.2 (0.62)

129. Secondary Outcome: Changes From Baseline to Week 24 in the Simpson-Angus Extrapyramidal Symptoms (EPS) Scale Total Score
Description: The Simpson-Angus EPS Scale is a clinician-rated scale to assess parkinsonian and extrapyramidal symptoms (10 items) associated with antipsychotic medications. Each item is rated on a 5-point scale. In addition, this scale was used to evaluate and characterize adverse events of extrapyramidal symptoms. Total scores are calculated by summing the scores of each item (minimum 0, maximum 40) and dividing by the number of items (10). Scores can range from 0-4. A higher score indicates more severe symptoms. Data represents change from baseline to week 24, positive values represent worsening.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
units on a scale | 0.0 (0.71) | 0.0 (0.53) | -0.1 (0.45) | -0.2 (0.58)

130. Secondary Outcome: Change From Baseline to Endpoint in the Barnes Akathisia Rating Scale (BARS) Total Score
Description: Barnes Akathisia Rating Scale (BARS) measures presence and severity of drug-induced akathisia. Items related to objective akathisia, subjective awareness of restlessness, and distress related to restlessness were rated using a 4-point scale: 0=normal/no distress, 1=presence of restlessness/mild distress, 2=observable restlessness/moderate distress, 3=constant restlessness/severe distress. Total score is sum of scores of each item and range from 0-9. Higher score indicates greater restlessness and distress. Data represent change from baseline to endpoint, positive values represent worsening.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
units on a scale | 0.0 (0.58) | -0.3 (1.03) | 0.0 (0.53) | -0.1 (0.69)

131. Secondary Outcome: Change From Baseline to Week 1 in the Barnes Akathisia Rating Scale (BARS) Total Score
Description: Barnes Akathisia Rating Scale (BARS) measures presence and severity of drug-induced akathisia. Items related to objective akathisia, subjective awareness of restlessness, and distress related to restlessness were rated using a 4-point scale: 0=normal/no distress, 1=presence of restlessness/mild distress, 2=observable restlessness/moderate distress, 3=constant restlessness/severe distress. Total score is sum of scores of each item and range from 0-9. Higher score indicates greater restlessness and distress. Data represent change from baseline to week 1, positive values represent worsening.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
units on a scale | 0.0 (0.55) | -0.3 (0.93) | 0.0 (0.30) | 0.1 (0.95)

132. Secondary Outcome: Change From Baseline to Week 2 in the Barnes Akathisia Rating Scale (BARS) Total Score
Description: Barnes Akathisia Rating Scale (BARS) measures presence and severity of drug-induced akathisia. Items related to objective akathisia, subjective awareness of restlessness, and distress related to restlessness were rated using a 4-point scale: 0=normal/no distress, 1=presence of restlessness/mild distress, 2=observable restlessness/moderate distress, 3=constant restlessness/severe distress. Total score is sum of scores of each item and range from 0-9. Higher score indicates greater restlessness and distress. Data represent change from baseline to week 2, positive values represent worsening.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
units on a scale | 0.0 (0.60) | -0.1 (1.07) | 0.1 (0.36) | 0.1 (0.93)

133. Secondary Outcome: Change From Baseline to Week 4 in the Barnes Akathisia Rating Scale (BARS) Total Score
Description: Barnes Akathisia Rating Scale (BARS) measures presence and severity of drug-induced akathisia. Items related to objective akathisia, subjective awareness of restlessness, and distress related to restlessness were rated using a 4-point scale: 0=normal/no distress, 1=presence of restlessness/mild distress, 2=observable restlessness/moderate distress, 3=constant restlessness/severe distress. Total score is sum of scores of each item and range from 0-9. Higher score indicates greater restlessness and distress. Data represent change from baseline to week 4, positive values represent worsening.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 62
units on a scale | 0.0 (0.60) | -0.2 (0.95) | 0.0 (0.33) | -0.1 (0.70)

134. Secondary Outcome: Change From Baseline to Week 8 in the Barnes Akathisia Rating Scale (BARS) Total Score
Description: Barnes Akathisia Rating Scale (BARS) measures presence and severity of drug-induced akathisia. Items related to objective akathisia, subjective awareness of restlessness, and distress related to restlessness were rated using a 4-point scale: 0=normal/no distress, 1=presence of restlessness/mild distress, 2=observable restlessness/moderate distress, 3=constant restlessness/severe distress. Total score is sum of scores of each item and range from 0-9. Higher score indicates greater restlessness and distress. Data represent change from baseline to week 8, positive values represent worsening.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 54
units on a scale | 0.0 (0.19) | -0.2 (0.98) | 0.1 (1.12) | 0.0 (1.57)

135. Secondary Outcome: Change From Baseline to Week 12 in the Barnes Akathisia Rating Scale (BARS) Total Score
Description: Barnes Akathisia Rating Scale (BARS) measures presence and severity of drug-induced akathisia. Items related to objective akathisia, subjective awareness of restlessness, and distress related to restlessness were rated using a 4-point scale: 0=normal/no distress, 1=presence of restlessness/mild distress, 2=observable restlessness/moderate distress, 3=constant restlessness/severe distress. Total score is sum of scores of each item and range from 0-9. Higher score indicates greater restlessness and distress. Data represent change from baseline to week 12, positive values represent worsening.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
units on a scale | 0.1 (0.33) | -0.4 (1.00) | 0.2 (1.34) | 0.0 (1.59)

136. Secondary Outcome: Change From Baseline to Week 16 in the Barnes Akathisia Rating Scale (BARS) Total Score
Description: Barnes Akathisia Rating Scale (BARS) measures presence and severity of drug-induced akathisia. Items related to objective akathisia, subjective awareness of restlessness, and distress related to restlessness were rated using a 4-point scale: 0=normal/no distress, 1=presence of restlessness/mild distress, 2=observable restlessness/moderate distress, 3=constant restlessness/severe distress. Total score is sum of scores of each item and range from 0-9. Higher score indicates greater restlessness and distress. Data represent change from baseline to week 16, positive values represent worsening.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
units on a scale | 0.1 (0.61) | -0.3 (0.83) | 0.1 (0.90) | -0.2 (0.95)

137. Secondary Outcome: Change From Baseline to Week 20 in the Barnes Akathisia Rating Scale (BARS) Total Score
Description: Barnes Akathisia Rating Scale (BARS) measures presence and severity of drug-induced akathisia. Items related to objective akathisia, subjective awareness of restlessness, and distress related to restlessness were rated using a 4-point scale: 0=normal/no distress, 1=presence of restlessness/mild distress, 2=observable restlessness/moderate distress, 3=constant restlessness/severe distress. Total score is sum of scores of each item and range from 0-9. Higher score indicates greater restlessness and distress. Data represent change from baseline to week 20, positive values represent worsening.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
units on a scale | 0.0 (0.14) | -0.2 (0.98) | 0.1 (1.06) | -0.3 (0.85)

138. Secondary Outcome: Change From Baseline to Week 24 in the Barnes Akathisia Rating Scale (BARS) Total Score
Description: Barnes Akathisia Rating Scale (BARS) measures presence and severity of drug-induced akathisia. Items related to objective akathisia, subjective awareness of restlessness, and distress related to restlessness were rated using a 4-point scale: 0=normal/no distress, 1=presence of restlessness/mild distress, 2=observable restlessness/moderate distress, 3=constant restlessness/severe distress. Total score is sum of scores of each item and range from 0-9. Higher score indicates greater restlessness and distress. Data represent change from baseline to week 24, positive values represent worsening.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
units on a scale | 0.1 (0.39) | -0.5 (1.11) | 0.0 (0.57) | -0.2 (0.76)

139. Secondary Outcome: Change From Baseline to Endpoint in the Calgary Depression Scale for Schizophrenia (CDSS) Score
Description: Calgary Depression Scale for Schizophrenia (CDSS) assesses the level of depression in patients with schizophrenia. Nine items (depression, hopelessness, self-depreciation, pathological guilt, guilty ideas of reference, morning depression, early awakening, suicidal, observed depression) are each scored on a 4-point scale: 0=absent, 1=mild, 2=moderate, 3=severe. The total score is a sum of the scores of each item and may range from 0 to 27. Higher score more severe pathology. Data presented here represents the change from baseline to endpoint, positive values represent worsening.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 70 | 69 | 71 | 70
units on a scale | -0.1 (2.24) | -0.6 (2.14) | 0.1 (2.80) | 0.1 (2.96)

140. Secondary Outcome: Change From Baseline to Week 1 in the Calgary Depression Scale for Schizophrenia (CDSS) Score
Description: Calgary Depression Scale for Schizophrenia (CDSS) assesses the level of depression in patients with schizophrenia. Nine items (depression, hopelessness, self-depreciation, pathological guilt, guilty ideas of reference, morning depression, early awakening, suicidal, observed depression) are each scored on a 4-point scale: 0=absent, 1=mild, 2=moderate, 3=severe. The total score is a sum of the scores of each item and may range from 0 to 27. Higher score more severe pathology. Data presented here represents the change from baseline to week 1, positive values represent worsening.
Time Frame: Baseline and Week 1
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 69 | 66 | 69 | 70
units on a scale | -0.3 (2.13) | -0.9 (1.68) | 0.2 (2.05) | -0.7 (2.44)

141. Secondary Outcome: Change From Baseline to Week 2 in the Calgary Depression Scale for Schizophrenia (CDSS) Score
Description: Calgary Depression Scale for Schizophrenia (CDSS) assesses the level of depression in patients with schizophrenia. Nine items (depression, hopelessness, self-depreciation, pathological guilt, guilty ideas of reference, morning depression, early awakening, suicidal, observed depression) are each scored on a 4-point scale: 0=absent, 1=mild, 2=moderate, 3=severe. The total score is a sum of the scores of each item and may range from 0 to 27. Higher score more severe pathology. Data presented here represents the change from baseline to week 2, positive values represent worsening.
Time Frame: Baseline and Week 2
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 65 | 63 | 68 | 66
units on a scale | -0.5 (1.77) | -0.7 (1.90) | -0.2 (1.77) | -0.7 (2.25)

142. Secondary Outcome: Change From Baseline to Week 4 in the Calgary Depression Scale for Schizophrenia (CDSS) Score
Description: Calgary Depression Scale for Schizophrenia (CDSS) assesses the level of depression in patients with schizophrenia. Nine items (depression, hopelessness, self-depreciation, pathological guilt, guilty ideas of reference, morning depression, early awakening, suicidal, observed depression) are each scored on a 4-point scale: 0=absent, 1=mild, 2=moderate, 3=severe. The total score is a sum of the scores of each item and may range from 0 to 27. Higher score more severe pathology. Data presented here represents the change from baseline to week 4, positive values represent worsening.
Time Frame: Baseline and Week 4
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 59 | 65 | 61
units on a scale | -0.3 (2.39) | -0.7 (1.70) | -0.5 (2.06) | -0.5 (2.71)

143. Secondary Outcome: Change From Baseline to Week 8 in the Calgary Depression Scale for Schizophrenia (CDSS) Score
Description: Calgary Depression Scale for Schizophrenia (CDSS) assesses the level of depression in patients with schizophrenia. Nine items (depression, hopelessness, self-depreciation, pathological guilt, guilty ideas of reference, morning depression, early awakening, suicidal, observed depression) are each scored on a 4-point scale: 0=absent, 1=mild, 2=moderate, 3=severe. The total score is a sum of the scores of each item and may range from 0 to 27. Higher score more severe pathology. Data presented here represents the change from baseline to week 8, positive values represent worsening.
Time Frame: Baseline and Week 8
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 55
units on a scale | -0.3 (2.09) | -0.6 (1.62) | -0.4 (2.22) | -0.6 (2.74)

144. Secondary Outcome: Change From Baseline to Week 12 in the Calgary Depression Scale for Schizophrenia (CDSS) Score
Description: Calgary Depression Scale for Schizophrenia (CDSS) assesses the level of depression in patients with schizophrenia. Nine items (depression, hopelessness, self-depreciation, pathological guilt, guilty ideas of reference, morning depression, early awakening, suicidal, observed depression) are each scored on a 4-point scale: 0=absent, 1=mild, 2=moderate, 3=severe. The total score is a sum of the scores of each item and may range from 0 to 27. Higher score more severe pathology. Data presented here represents the change from baseline to week 12, positive values represent worsening.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 51 | 49 | 53 | 51
units on a scale | 0.3 (2.49) | -0.9 (1.55) | -0.1 (2.42) | -0.4 (2.39)

145. Secondary Outcome: Change From Baseline to Week 16 in the Calgary Depression Scale for Schizophrenia (CDSS) Score
Description: Calgary Depression Scale for Schizophrenia (CDSS) assesses the level of depression in patients with schizophrenia. Nine items (depression, hopelessness, self-depreciation, pathological guilt, guilty ideas of reference, morning depression, early awakening, suicidal, observed depression) are each scored on a 4-point scale: 0=absent, 1=mild, 2=moderate, 3=severe. The total score is a sum of the scores of each item and may range from 0 to 27. Higher score more severe pathology. Data presented here represents the change from baseline to week 16, positive values represent worsening.
Time Frame: Baseline and Week 16
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 50 | 43 | 49 | 49
units on a scale | 0.0 (2.74) | -0.7 (1.95) | -0.6 (2.13) | -0.2 (2.06)

146. Secondary Outcome: Change From Baseline to Week 20 in the Calgary Depression Scale for Schizophrenia (CDSS) Score
Description: Calgary Depression Scale for Schizophrenia (CDSS) assesses the level of depression in patients with schizophrenia. Nine items (depression, hopelessness, self-depreciation, pathological guilt, guilty ideas of reference, morning depression, early awakening, suicidal, observed depression) are each scored on a 4-point scale: 0=absent, 1=mild, 2=moderate, 3=severe. The total score is a sum of the scores of each item and may range from 0 to 27. Higher score more severe pathology. Data presented here represents the change from baseline to week 20, positive values represent worsening.
Time Frame: Baseline and Week 20
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 49 | 42 | 45 | 47
units on a scale | -0.2 (2.67) | -0.5 (1.69) | -0.4 (2.67) | -0.8 (2.09)

147. Secondary Outcome: Change From Baseline to Week 24 in the Calgary Depression Scale for Schizophrenia (CDSS) Score
Description: Calgary Depression Scale for Schizophrenia (CDSS) assesses the level of depression in patients with schizophrenia. Nine items (depression, hopelessness, self-depreciation, pathological guilt, guilty ideas of reference, morning depression, early awakening, suicidal, observed depression) are each scored on a 4-point scale: 0=absent, 1=mild, 2=moderate, 3=severe. The total score is a sum of the scores of each item and may range from 0 to 27. Higher score more severe pathology. Data presented here represents the change from baseline to week 24, positive values represent worsening.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
units on a scale | 0.1 (2.32) | -1.0 (1.83) | -0.1 (2.71) | -0.6 (2.81)

148. Secondary Outcome: Columbia Suicide-Severity Rating Scale (C-SSRS) Scores - Percentage of Participants With Suicidal Behavior at Endpoint
Description: The C-SSRS was performed at weeks 8, 16, and 24 (or last observation after baseline), and at any time if clinically indicated. The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The data presented here represents the percentage of patients in each arm found to have suicidal behavior in the judgment of a clinician and based upon a clinicians interpretation of the subject's responses to the C-SSRS questions.
Time Frame: Endpoint (Week 24 or last observation)
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 71 | 69 | 71 | 70
Percentage of participants | 1 | 0 | 0 | 0

149. Secondary Outcome: Columbia Suicide-Severity Rating Scale (C-SSRS) Scores - Percentage of Participants With Suicidal Behavior at Week 8
Description: The C-SSRS was performed at weeks 8, 16, and 24 (or last observation after baseline), and at any time if clinically indicated. The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The data presented here represents the percentage of patients in each arm found to have suicidal behavior at week 8 in the judgment of a clinician and based upon a clinicians interpretation of the subject's responses to the C-SSRS questions.
Time Frame: Week 8
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 71 | 69 | 71 | 70
Percentage of participants | 0 | 0 | 0 | 0

150. Secondary Outcome: Columbia Suicide-Severity Rating Scale (C-SSRS) Scores - Percentage of Participants With Suicidal Behavior at Week 16
Description: The C-SSRS was performed at weeks 8, 16, and 24 (or last observation after baseline), and at any time if clinically indicated. The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The data presented here represents the percentage of patients in each arm found to have suicidal behavior in the judgment of a clinician and based upon a clinicians interpretation of the subject's responses to the C-SSRS questions at week 16.
Time Frame: Week 16
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 71 | 69 | 71 | 70
Percentage of participants | 0 | 0 | 0 | 1

151. Secondary Outcome: Columbia Suicide-Severity Rating Scale (C-SSRS) Scores - Percentage of Participants With Suicidal Behavior at Week 24
Description: The C-SSRS was performed at weeks 8, 16, and 24 (or last observation after baseline), and at any time if clinically indicated. The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The data presented here represents the percentage of patients in each arm found to have suicidal behavior in the judgment of a clinician and based upon a clinicians interpretation of the subject's responses to the C-SSRS questions at week 24.
Time Frame: Week 24
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 71 | 69 | 71 | 70
Percentage of participants | 0 | 0 | 0 | 0

152. Secondary Outcome: Columbia Suicide-Severity Rating Scale (C-SSRS) Scores - Percentage of Participants With Suicidal Ideations at Endpoint
Description: The C-SSRS was performed at weeks 8, 16, and 24 (or last observation after baseline), and at any time if clinically indicated. The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The data presented here represents the percentage of patients in each arm found to have suicidal ideation in the judgment of a clinician and based upon a clinicians interpretation of the subject's responses to the C-SSRS questions at endpoint.
Time Frame: Endpoint (Week 24 or last observation)
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 71 | 69 | 71 | 70
Percentage of participants | 1 | 1 | 4 | 3

153. Secondary Outcome: Columbia Suicide-Severity Rating Scale (C-SSRS) Scores - Percentage of Participants With Suicidal Ideations at Week 8
Description: The C-SSRS was performed at weeks 8, 16, and 24 (or last observation after baseline), and at any time if clinically indicated. The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The data presented here represents the percentage of patients in each arm found to have suicidal ideation in the judgment of a clinician and based upon a clinicians interpretation of the subject's responses to the C-SSRS questions at week 8.
Time Frame: Week 8
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 71 | 69 | 71 | 70
Percentage of participants | 1 | 0 | 1 | 0

154. Secondary Outcome: Columbia Suicide-Severity Rating Scale (C-SSRS) Scores - Percentage of Participants With Suicidal Ideations at Week 16
Description: The C-SSRS was performed at weeks 8, 16, and 24 (or last observation after baseline), and at any time if clinically indicated. The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The data presented here represents the percentage of patients in each arm found to have suicidal ideation in the judgment of a clinician and based upon a clinicians interpretation of the subject's responses to the C-SSRS questions at week 16.
Time Frame: Week 16
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 71 | 69 | 71 | 70
percentage of participants | 0 | 0 | 1 | 1

155. Secondary Outcome: Columbia Suicide-Severity Rating Scale (C-SSRS) Scores - Percentage of Participants With Suicidal Ideations at Week 24
Description: The C-SSRS was performed at weeks 8, 16, and 24 (or last observation after baseline), and at any time if clinically indicated. The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The data presented here represents the percentage of patients in each arm found to have suicidal ideation in the judgment of a clinician and based upon a clinicians interpretation of the subject's responses to the C-SSRS questions at week 24.
Time Frame: Week 24
Population: The number of participants analyzed represents the number of participants with evaluable data.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 71 | 69 | 71 | 70
Percentage of participants | 0 | 0 | 3 | 0

156. Secondary Outcome: Change From Baseline to Endpoint in Sleep Latency
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency (time till fall asleep), duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to endpoint in reported sleep latency. There is no range of possible values, positive values represent prolongation of sleep latency.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 69 | 62 | 68
Minutes | 2.0 (39.33) | -8.2 (39.42) | -1.5 (38.98) | -1.2 (33.80)

157. Secondary Outcome: Change From Baseline to Week 12 in Sleep Latency
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency (time till fall asleep), duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to week 12 in reported sleep latency. There is no range of possible values, positive values represent prolongation of sleep latency.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Minutes | -0.6 (36.91) | -5.6 (43.19) | -2.6 (46.64) | -2.5 (30.12)

158. Secondary Outcome: Change From Baseline to Week 24 in Sleep Latency
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency (time till fall asleep), duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to week 24 in reported sleep latency. There is no range of possible values, positive values represent prolongation of sleep latency.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 45 | 40 | 44 | 46
Minutes | -2.4 (30.87) | -5.4 (44.89) | -7.3 (39.53) | -4.4 (31.80)

159. Secondary Outcome: Change From Baseline to Endpoint in Number of Nighttime Awakenings
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to endpoint in reported number of nighttime awakenings. A positive value represents an increase in number of night time awakenings.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Awakenings
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 69 | 62 | 68
Awakenings | 0.1 (1.91) | 0.0 (2.07) | -0.1 (1.32) | -0.6 (1.91)

160. Secondary Outcome: Change From Baseline to Week 12 in Number of Nighttime Awakenings
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to week 12 in reported number of nighttime awakenings. A positive value represents an increase in number of night time awakenings.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Awakenings
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Awakenings | -0.2 (1.32) | -0.3 (1.49) | -0.1 (1.33) | -0.1 (1.59)

161. Secondary Outcome: Change From Baseline to Week 24 in Number of Nighttime Awakenings
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to week 24 in reported number of nighttime awakenings. A positive value represents an increase in number of night time awakenings.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Awakenings
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 45 | 40 | 44 | 46
Awakenings | 0.2 (2.19) | -0.2 (1.67) | 0.0 (1.36) | -0.5 (1.70)

162. Secondary Outcome: Change From Baseline to Endpoint in Time Spent Awake at Night
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to endpoint in reported time spent awake at night. A positive value represents longer period awake at night.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 69 | 62 | 68
Minutes | -2.7 (36.34) | -1.8 (45.40) | -0.2 (43.96) | 3.2 (34.01)

163. Secondary Outcome: Change From Baseline to Week 12 in Time Spent Awake at Night
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to week 12 in reported time spent awake at night. A positive value represents longer period awake at night.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Minutes | -2.6 (28.59) | -4.7 (31.47) | 0.2 (39.32) | -0.3 (29.21)

164. Secondary Outcome: Change From Baseline to Week 24 in Time Spent Awake at Night
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to week 24 in reported time spent awake at night. A positive value represents longer period awake at night.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 45 | 40 | 44 | 46
Minutes | -4.1 (41.62) | -1.8 (47.46) | -2.4 (36.56) | -1.8 (28.58)

165. Secondary Outcome: Change From Baseline to Endpoint in Time Spent Asleep at Night
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to endpoint in reported time spent asleep at night. A positive value indicates increased time spent asleep at night.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 62 | 69 | 62 | 68
Minutes | -23.7 (115.55) | -20.1 (86.21) | -0.7 (91.18) | 5.3 (87.84)

166. Secondary Outcome: Change From Baseline to Week 12 in Time Spent Asleep at Night
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to week 12 in reported time spent asleep at night. A positive value indicates increased time spent asleep at night.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
Minutes | -12.7 (95.69) | -2.2 (115.90) | 10.9 (111.03) | 13.6 (102.58)

167. Secondary Outcome: Change From Baseline to Week 24 in Time Spent Asleep at Night
Description: A sleep questionnaire was used to evaluate the effect of armodafinil treatment on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to week 24 in reported time spent asleep at night. A positive value indicates increased time spent asleep at night.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 45 | 40 | 44 | 46
Minutes | -7.9 (121.18) | -22.4 (91.71) | 9.4 (88.00) | 9.6 (86.92)

168. Secondary Outcome: Change From Baseline to Endpoint in Sleep Quality Rating
Description: A sleep questionnaire was used to evaluate the effect of armodafinil on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to endpoint in participants' ratings of their quality of sleep as measured on a 4-point scale (1=Poor, 2=Fair, 3=Good, 4=Excellent). A positive value represents improvement in sleep quality.
Time Frame: Baseline and Endpoint (Week 24 or last observation)
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 63 | 69 | 62 | 68
units on a scale | 0.1 (0.78) | -0.1 (0.85) | -0.1 (0.83) | -0.1 (0.77)

169. Secondary Outcome: Change From Baseline to Week 12 in Sleep Quality Rating
Description: A sleep questionnaire was used to evaluate the effect of armodafinil on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to week 12 in participants' ratings of their quality of sleep as measured on a 4-point scale (1=Poor, 2=Fair, 3=Good, 4=Excellent). A positive value represents improvement in sleep quality.
Time Frame: Baseline and Week 12
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 52 | 49 | 53 | 51
units on a scale | -0.1 (0.71) | 0.0 (0.84) | -0.2 (0.89) | -0.2 (0.83)

170. Secondary Outcome: Change From Baseline to Week 24 in Sleep Quality Rating
Description: A sleep questionnaire was used to evaluate the effect of armodafinil on the patient's nighttime sleep. Patients completed the questionnaire to evaluate the sleep latency, duration, nighttime awakenings, and overall sleep quality. The questionnaire was assessed at the screening visit and at weeks 12 and 24 (or last visit after baseline). The data presented here represents the change from baseline to week 24 in participants' ratings of their quality of sleep as measured on a 4-point scale (1=Poor, 2=Fair, 3=Good, 4=Excellent). A positive value represents improvement in sleep quality.
Time Frame: Baseline and Week 24
Population: The number of participants with evaluable data (who completed the assessments at baseline and endpoint) are presented.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Number analyzed (Participants) | 46 | 40 | 44 | 46
Units on a scale | 0.0 (0.83) | 0.0 (0.86) | -0.2 (0.73) | -0.3 (0.65)

ADVERSE EVENTS:
Time Frame: The study period was defined as that time period from signature of the informed consent form through the end of the follow-up period. For this study, the follow-up period was defined as 7±2 days after the last dose of study drug.
Description: During each contact with the patient, the investigator queried the patient for adverse events by asking an open-ended question such as, "Have you had any unusual symptoms or medical problems since the last visit? If yes, please describe."
Arm/Group | 150 mg/Day Armodafinil | 200 mg/Day Armodafinil | 250 mg/Day Armodafinil | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 4/71 | 5/69 | 3/71 | 5/70
Other Adverse Events (participants affected / at risk) | 32/71 | 30/69 | 38/71 | 33/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 150 mg/Day Armodafinil (N=71) | 200 mg/Day Armodafinil (N=69) | 250 mg/Day Armodafinil (N=71) | Matching Placebo (N=70)
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 2 | 2 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Social stay hospitalisation (Social circumstances) | 0 | 0 | 0 | 2
Knee operation (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 150 mg/Day Armodafinil (N=71) | 200 mg/Day Armodafinil (N=69) | 250 mg/Day Armodafinil (N=71) | Matching Placebo (N=70)
Nausea (Gastrointestinal disorders) | 3 | 7 | 5 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 3 | 6 | 3
Toothache (Gastrointestinal disorders) | 3 | 3 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 4 | 5
Weight increased (Investigations) | 5 | 4 | 5 | 6
Headache (Nervous system disorders) | 10 | 7 | 14 | 6
Dizziness (Nervous system disorders) | 5 | 3 | 2 | 6
Initial insomnia (Psychiatric disorders) | 7 | 3 | 9 | 1
Anxiety (Psychiatric disorders) | 3 | 3 | 5 | 10
Schizophrenia (Psychiatric disorders) | 3 | 4 | 2 | 3
Suicidal ideation (Psychiatric disorders) | 2 | 1 | 5 | 3
Agitation (Psychiatric disorders) | 1 | 4 | 2 | 0
Psychotic disorder (Psychiatric disorders) | 3 | 2 | 1 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days